CLINICAL TRIAL: NCT02120352
Title: A Phase IIb Study Evaluating a Long-Acting Intramuscular Regimen of GSK1265744 Plus TMC278 For The Maintenance of Virologic Suppression Following an Induction of Virologic Suppression on an Oral Regimen of GSK1265744 Plus Abacavir/Lamivudine in HIV-1 Infected, Antiretroviral Therapy-Naive Adult Subjects
Brief Title: A Phase IIb Study to Evaluate a Long-Acting Intramuscular Regimen for Maintenance of Virologic Suppression (Following Induction With an Oral Regimen of GSK1265744 and Abacavir/Lamivudine) in Human Immunodeficiency Virus Type 1 (HIV-1) Infected, Antiretroviral Therapy-Naive Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200056; 2013-000783-29 (EudraCT Number)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: bi-monthly; GSK744; injectable; long acting; maintenance; abacavir; every other month; rilpivirine; HIV-1 infection; integrase inhibitor; TMC278 LA; RPV; non-nucleoside reverse transcriptase inhibitor; LA; once monthly; GSK1265744; induction; treatment satisfication; once daily; lamivudine; adherence; TMC278; therapy-naive
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) (Experimental): On Day 1 of the Maintenance period, participants who successfully completed the Induction period, were randomized to receive following intramuscular (IM) doses: Day 1 only: CAB long acting (LA) 800 mg (loading dose delivered as two 400 mg IM injections) + RPV LA 900 mg IM; Week 4 only: CAB LA 600 mg IM (second loading dose, no RPV); and from Week 8: CAB LA 600 mg IM +RPV LA 900 mg IM every 8 Weeks (Q8W) for 96 weeks. Eligible participants had the option to continue study participation in the Extension Period.
  Interventions: Drug: CAB LA; Drug: RPV
- CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) (Experimental): On Day 1 of the Maintenance period, participants who successfully completed the Induction period, were randomized to receive following IM doses: Day 1 only: CAB LA 800 mg (loading dose delivered as two 400 mg IM injections) + RPV LA 600 mg IM; and from Week 4: CAB LA 400 mg IM + RPV LA 600 mg IM every 4 Weeks (Q4W) for 96 weeks. Eligible participants had the option to continue study participation in the Extension Period.
  Interventions: Drug: CAB LA; Drug: RPV
- CAB 30 mg+ABC/3TC QD (Induction Period) (Active Comparator): In induction period, all participants received an oral regimen of cabotegravir (CAB) 30 milligrams (mg) once daily (QD) plus abacavir/lamivudine (ABC/3TC) 600/300 mg QD for 20 weeks. They also received an oral dose of Rilpivirine (RPV) 25 mg tablet once daily in the last 4 weeks of the Induction Period.
  Interventions: Drug: CAB Oral Tablets; Drug: ABC/3TC Oral tablets; Drug: RPV Oral Tablets
- CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period) (Active Comparator): On Day 1 of the Maintenance period, participants who successfully completed the Induction period, were randomized to receive CAB and ABC/3TC QD for 96 weeks. Eligible participants had the option to continue study participation in Extension Period by switching to an optimized IM CAB LA+ RPV LA regimen of their choice (Q8W or Q4W).
  Interventions: Drug: CAB Oral Tablets; Drug: ABC/3TC Oral tablets; Drug: RPV Oral Tablets
- Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) (Experimental): Participants who completed 96 weeks of CAB 30 mg + ABC/3TC QD regimen in Maintenance Period transitioned to Extension Period and received an optimized loading dose of CAB LA 600 mg+RPV LA 900 mg IM at Week 100 and Week 104 followed by CAB LA 600 mg+RPV LA 900 mg IM-Q8W in the Extension Phase. Participants were followed up until end of Extension Period.
  Interventions: Drug: CAB LA; Drug: RPV
- Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) (Experimental): Participants who completed 96 weeks of CAB 30 mg + ABC/3TC QD regimen in Maintenance Period transitioned to Extension Period and received an optimized loading dose of CAB LA 400 mg+RPV LA 900 mg IM at Week 100 followed by CAB LA 400 mg+RPV LA 900 mg IM-Q8W in the Extension Phase. Participants were followed up until end of Extension Period.
  Interventions: Drug: CAB LA; Drug: RPV
- Long-Term Follow-Up Group (Other): This group included participants that were withdrawn from CAB LA+RPV LA IM regimens based on protocol criteria and were required to access Highly Active Antiretroviral Therapy (HAART) of choice. Participants were followed up for approximately 52 weeks.
  Interventions: Other: HAART

INTERVENTIONS:
Drug: CAB Oral Tablets — White to almost white oval shaped film coated 30 mg tablets for oral administration.
  Arms: CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period); CAB 30 mg+ABC/3TC QD (Induction Period)
Drug: CAB LA — Sterile white to slightly colored suspension containing 200 mg/mL of GSK744 as free acid (GSK1265744 free acid), polysorbate 20, polyethylene glycol 3350, mannitol, and water for injection, packaged in a 3 mL USP Type I glass vial, for administration by IM injection
  Arms: CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period); CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period); Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period); Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period)
Drug: ABC/3TC Oral tablets — ABC/3TC fixed dose combination (FDC) oral tablet, containing 600 mg of ABC (as abacavir sulfate) and 300 mg of 3TC
  Arms: CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period); CAB 30 mg+ABC/3TC QD (Induction Period)
Drug: RPV Oral Tablets — Off-white, round, biconvex, film-coated 25 mg Rilpivirine (RPV) tablets for oral administration. Eligible subjects switching from the oral regimen to the IM regimen in the Extension Period will receive 2 weeks of RPV 25 mg once daily, from Week 102 through Week 104
  Arms: CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period); CAB 30 mg+ABC/3TC QD (Induction Period)
Other: HAART — Higly-active antiretroviral therapy chosen by participant based on investigator recommendations and based on availability.
  Arms: Long-Term Follow-Up Group
Drug: RPV — Sterile white suspension containing 300 mg/mL of TMC278 as free base, poloxamer 338, sodium dihydrogen phosphate monohydrate, citric acid monohydrate, glucose monohydrate, sodium hydroxide, water for injection, packaged in a 2 mL USP Type I glass vial, for administration by IM injection.
  Arms: CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period); CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period); Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period); Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period)

SUMMARY:
This study is a Phase IIb, randomized, multicentre, parallel group, open-label, study having an overall objective to evaluate the antiviral activity, tolerability, and safety of two intramuscular (IM) dosing regimens of GSK744 LA plus TMC278 LA, relative to GSK744 30 milligram (mg) plus Abacavir/Lamivudine (ABC/3TC) given orally once daily (QD), in HIV-1 infected antiretroviral-naïve subjects. GSK744 is the oral formulation of GSK1265744 (cabotegravir), GSK744 LA is the long acting injectable formulation of GSK1265744 and TMC278 LA is the long acting injectable formulation of TMC278.

The study will consist of three parts: an Induction Period, Maintenance Period and Extension Period. There is also a Long-Term Follow Up Period for subjects who withdraw from the study and have received at least one dose of GSK744 LA and / or TMC278 LA. In the Induction Period, eligible subjects will receive a combination of an oral regimen of 30 mg of GSK744 and 600/300 mg of ABC/3TC, once daily for 20 weeks. In the Maintenance Period, eligible subjects will be randomized 2:2:1 at Day 1 to receive an IM regimen of GSK744 LA 400 mg + TMC278 LA 600 mg every 4 weeks for 96 weeks (Q4W), an IM regimen of GSK744 LA 600 mg + TMC278 LA 900 mg every 8 weeks for 96 weeks (Q8W), or to continue on the oral Induction Period regimen of GSK744 30 mg + ABC/3TC once daily for 96 weeks (or 104 weeks if continuing on to the Extension Period). The Extension Period will allow for a collection of longer term efficacy and safety and tolerability data from subjects receiving GSK744 LA and TMC278 LA.

The study will involve sufficient subjects at screening in order to ensure a total of approximately 265 subjects at the beginning of the Induction Period and approximately 225 subjects randomized into the Maintenance Period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects screened for this study must be HIV-1 infected and >=18 years of age.
* A female subject is eligible to enter and participate in the study if she: is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or; is of child-bearing potential with a negative pregnancy test at both Screening and first day of the Induction Period and agrees to use one of the following methods of contraception to avoid pregnancy 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all oral study medications and for at least 52 weeks after discontinuation of GSK744 LA and TMC278 LA: Complete abstinence from intercourse (where this is the subject's preferred and usual lifestyle); double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide); approved hormonal contraception; any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year; male partner sterilization prior to the female subject's entry into the study, and this male is the sole partner for that subject; any other method with published data showing that the lowest expected failure rate is <1% per year; any contraception method must be used consistently and in accordance with the approved product label. All subjects participating in the study must follow safer sexual practices including the use of effective barrier methods (e.g. male condom/spermicide) to minimize risk of HIV transmission.
* HIV-1 infection as documented by Screening plasma HIV-1 RNA>=1000 c/mL.
* CD4+ cell count >=200 cells/mm^3 (or higher as local guidelines dictate).
* ART-naive defined as having no more than 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection. Any previous exposure to an HIV integrase inhibitor or non-nucleoside reverse transcriptase inhibitor will be exclusionary.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Women who are breastfeeding.
* Any evidence at screening of an active Center for Disease and Prevention Control (CDC) Category C disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Subjects with known moderate to severe hepatic impairment.
* Any pre-existing physical or mental condition (including substance abuse disorder) which, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the subject.
* Subject who, in the investigator's judgment, poses a significant suicide risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk.
* The subject has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* History of ongoing or clinically relevant hepatitis within the previous 6 months, including chronic Hepatitis B virus (HBV) infection (HBsAg positive). Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; subjects who are anticipated to require such therapy during the randomized portion of the study must be excluded.
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* History of the following cardiac diseases: myocardial infarction, congestive heart failure, documented hypertrophic cardiomyopathy, sustained ventricular tachycardia.
* Personal or known family history of prolonged QT syndrome.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug or render the subject unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation.
* Any evidence of primary resistance based on the presence of any major resistance-associated mutation in the Screening result or, if known, any historical resistance test result.
* Any verified Grade 4 laboratory abnormality.
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound.
* Subject has estimated creatinine clearance <50 mL/min via Cockcroft-Gault method.
* Alanine aminotransferase (ALT) >=5 times Upper limit of normal (ULN). Subjects with ALT >2xULN but <5xULN may participate in the study, if in the opinion of the Investigator and GlaxoSmithKline (GSK) medical monitor the lab abnormality will not interfere with the study procedures or compromise subject safety.
* Alanine aminotransferase (ALT) >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin).
* Any clinically significant finding on screening or Baseline electrocardiograph (ECG), specifically: Heart rate <45 and >100 beats per minute (bpm) (Males) and <50 and >100 bpm (Females) (100 to 110 bpm can be rechecked within 30 minutes to verify eligibility), QRS duration >120 milliseconds (msec), QTc interval (B or F) >450 msec; non-sustained (>=3 consecutive beats) or sustained ventricular tachycardia; sinus pauses >2.5 seconds; 2nd degree (Type II) or higher atrio-ventricular (AV) block; evidence of WPW (Wolff- Parkinson-White) syndrome (ventricular pre-excitation); pathologic Q waves defined as Q wave >40msec OR depth >0.4 mV; any significant arrhythmia (either on ECG or by history) which, in the opinion of the Investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Subjects who are human leukocyte antigen (HLA)-B*5701 positive and unable to use an alternative nucleoside reverse transcriptase inhibitor (NRTI) backbone (subjects who are HLA-B*5701 positive may be enrolled if they use an alternative NRTI backbone that does not contain abacavir).
* Exposure to an experimental drug and/or experimental vaccine within 28 days or 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP.
* Treatment with any of the following agents within 28 days of Screening; radiation therapy, cytotoxic chemotherapeutic agents, tuberculosis therapy and Immunomodulators that alter immune responses (such as systemic corticosteroids, interleukins, or interferons)
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of the first dose of IP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2015-08-13 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (37):
- United States (15):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
- Canada (5):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
- Germany (6):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Kerrigan D, Mantsios A, Gorgolas M, Montes ML, Pulido F, Brinson C, deVente J, Richmond GJ, Beckham SW, Hammond P, Margolis D, Murray M. Experiences with long acting injectable ART: A qualitative study among PLHIV participating in a Phase II study of cabotegravir + rilpivirine (LATTE-2) in the United States and Spain. PLoS One. 2018 Jan 5;13(1):e0190487. doi: 10.1371/journal.pone.0190487. eCollection 2018. PMID 29304154
- [Derived] Okesanya OJ, Ayeni RA, Amadin P, Ngwoke I, Amisu BO, Ukoaka BM, Ahmed MM, Oso TA, Musa SS, Lucero-Prisno DE. Advances in HIV Treatment and Vaccine Development: Emerging Therapies and Breakthrough Strategies for Long-Term Control. AIDS Res Treat. 2025 Jul 4;2025:6829446. doi: 10.1155/arat/6829446. eCollection 2025. PMID 40655875
- [Derived] Smith GHR, Henry WK, Podzamczer D, Masia MDM, Bettacchi CJ, Arasteh K, Jaeger H, Khuong-Josses MA, Montes-Ramirez ML, Stellbrink HJ, Yazdanpanah Y, Richmond GJ, Sutton KC, Zhang F, McCoig CC, St Clair MH, Vandermeulen K, Van Solingen-Ristea R, Smith KY, Margolis DA, Spreen WR. Efficacy, Safety, and Durability of Long-Acting Cabotegravir and Rilpivirine in Adults With Human Immunodeficiency Virus Type 1 Infection: 5-Year Results From the LATTE-2 Study. Open Forum Infect Dis. 2021 Aug 25;8(9):ofab439. doi: 10.1093/ofid/ofab439. eCollection 2021 Sep. PMID 34557563
- [Derived] Letendre SL, Mills A, Hagins D, Swindells S, Felizarta F, Devente J, Bettacchi C, Lou Y, Ford S, Sutton K, Shaik JS, Crauwels H, D'Amico R, Patel P. Pharmacokinetics and antiviral activity of cabotegravir and rilpivirine in cerebrospinal fluid following long-acting injectable administration in HIV-infected adults. J Antimicrob Chemother. 2020 Mar 1;75(3):648-655. doi: 10.1093/jac/dkz504. PMID 31873746
- [Derived] Murray M, Pulido F, Mills A, Ramgopal M, LeBlanc R, Jaeger H, Canon V, Dorey D, Griffith S, Mrus J, Spreen W, Margolis D. Patient-reported tolerability and acceptability of cabotegravir + rilpivirine long-acting injections for the treatment of HIV-1 infection: 96-week results from the randomized LATTE-2 study. HIV Res Clin Pract. 2019 Aug-Oct;20(4-5):111-122. doi: 10.1080/25787489.2019.1661696. Epub 2019 Sep 18. PMID 31533539
- [Derived] Margolis DA, Gonzalez-Garcia J, Stellbrink HJ, Eron JJ, Yazdanpanah Y, Podzamczer D, Lutz T, Angel JB, Richmond GJ, Clotet B, Gutierrez F, Sloan L, Clair MS, Murray M, Ford SL, Mrus J, Patel P, Crauwels H, Griffith SK, Sutton KC, Dorey D, Smith KY, Williams PE, Spreen WR. Long-acting intramuscular cabotegravir and rilpivirine in adults with HIV-1 infection (LATTE-2): 96-week results of a randomised, open-label, phase 2b, non-inferiority trial. Lancet. 2017 Sep 23;390(10101):1499-1510. doi: 10.1016/S0140-6736(17)31917-7. Epub 2017 Jul 24. PMID 28750935

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 50 sites in five countries (United States, Canada, France, Germany and Spain). The results presented are based on final analysis, up to approximately Week 468.
Pre-assignment Details: Study consisted of 28 days Screening Period, 20 weeks Induction Period, 96 weeks Maintenance Period (MP), Extension Period (EP) and 52 weeks Long-Term Follow Up Period (LTFP). A total of 309 participants were enrolled in the study and entered the Induction Period, of which 288 completed and 286 were qualified and randomized into the MP.
Period: Induction Period (20 Weeks)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) | Long-Term Follow-Up Group
Started | 309 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 288 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 21 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Met protocol-defined stopping criteria | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (Up to Week 96)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) | Long-Term Follow-Up Group
Started (2 participants did not enter Maintenance phase as they had Day 1 viral loads >50 copies/milliliter.) | 0 | 115 | 115 | 56 | 0 | 0 | 0
Completed | 0 | 110 | 101 | 47 | 0 | 0 | 0
Not Completed | 0 | 5 | 14 | 9 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 8 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Met protocol-defined stopping criteria | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Extension Period (Week 97 to Study End)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) | Long-Term Follow-Up Group
Started | 0 | 107 | 101 | 0 | 34 | 10 | 0
Completed | 0 | 92 | 76 | 0 | 26 | 8 | 0
Not Completed | 0 | 15 | 25 | 0 | 8 | 2 | 0
Not completed — Adverse Event | 0 | 3 | 11 | 0 | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 9 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Site closed | 0 | 0 | 1 | 0 | 0 | 1 | 0
Period: Long-Term Follow-up Period (52 Weeks)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) | Long-Term Follow-Up Group
Started | 0 | 0 | 0 | 0 | 0 | 0 | 43
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: 309 participants are valid only for the Induction Phase of the study (Weeks -20 to Day 1). Participants (n=286) were randomized at Day 1 of the Maintenance Phase.
Groups:
- CAB 30 mg+ABC/3TC QD: In induction period, all participants received an oral regimen of cabotegravir (CAB) 30 milligrams (mg) once daily (QD) plus abacavir/lamivudine (ABC/3TC) 600/300 mg QD for 20 weeks. They also received an oral dose of Rilpivirine (RPV) 25 mg tablet once daily in the last 4 weeks of the Induction Period.
Arm/Group | CAB 30 mg+ABC/3TC QD
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American/African Heritage | 46
  Race: American Indian or Alaskan Native | 10
  Race: Asian - Central/South Asian Heritage | 1
  Race: Asian - Japanese Heritage | 1
  Race: Asian - South East Asian Heritage | 2
  Race: Native Hawaiian or Other Pacific Islander | 1
  Race: White - Arabic/North African Heritage | 6
  Race: White - White/Caucasian/European Heritage | 240
  Race: Mixed Race | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) Level Below 50 Copies/Milliliter (c/mL) at Week 32
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using Food and Drug Administration (FDA) Snapshot algorithm. The algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as well as participants who switch their concomitant antiretroviral therapy (ART) prior to the visit of interest as non-responders. The Intent-to-Treat Maintenance Exposed (ITT-ME) Population consisted of all randomized participants who received at least one injection or one dose of investigational product during the Maintenance Period of the study (on or after Day 1 visit).
Time Frame: Week 32
Population: ITT-ME Population
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Percentage of participants | 95 | 94 | 91
Statistical Analysis 1: Comparison: CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) vs CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period); Test type: Other; Difference in Percentage = 3.7, 95% CI 2-sided [-4.8 to 12.2] — Comparison between CAB LA 600 mg+RPV LA 900 mg IM-Q8W and CAB 30 mg+ABC/3TC QD
Statistical Analysis 2: Comparison: CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) vs CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period); Test type: Other; Difference in Percentage = 2.8, 95% CI 2-sided [-5.8 to 11.5] — Comparison between CAB LA 400 mg+RPV LA 600 mg IM-Q4W and CAB 30 mg+ABC/3TC QD

2. Primary Outcome: Number of Participants With Protocol Defined Virologic Failure (PDVF) Until Week 32
Description: Virologic failure was defined as any of the following: (1) Non-response as indicated by a less than 1.0 logarithm to base 10 (log10) c/mL decrease in plasma HIV-1 RNA after 4 weeks of starting the Induction Period, which is subsequently confirmed, unless the plasma HIV-1 RNA is < 400 c/mL; (2) Rebound as indicated by two consecutive plasma HIV-1 RNA levels >=200 c/mL after prior suppression to < 200 c/mL; (3) Rebound as indicated by two consecutive plasma HIV-1 RNA that are > 0.5 log10 c/mL increase in plasma HIV-1 RNA from the nadir value on study, where the lowest HIV-1 RNA value is >=200 c/mL.
Time Frame: Up to Week 32
Population: ITT-ME Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants | 1 | 0 | 1

3. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event (Non-SAE) (Induction Period)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, important medical events which may require medical or surgical intervention, drug-induced liver injury with hyperbilirubinaemia.
Time Frame: Up to 20 weeks
Population: Safety Population. It consists of all enrolled subjects who received at least one dose of investigational product during induction period.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Participants
  Any non-SAE | 246
  Any SAE | 8

4. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Any Non-serious Adverse Event (Non-SAE) (Maintenance Period)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, important medical events which may require medical or surgical intervention, drug-induced liver injury with hyperbilirubinaemia. Data presented includes all post-baseline induction period and maintenance period adverse events, as well as long-term follow-up period adverse events for those participants who did not enter the extension period.
Time Frame: Up to an average of 59 weeks
Population: Safety Maintenance Population. It consisted of all participants who entered the Maintenance period and received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Any non-SAE | 115 | 113 | 52
  Any SAE | 9 | 8 | 5

5. Primary Outcome: Number of Participants With Post-Baseline Adverse Events by Maximum Toxicity Grade
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Toxicity was graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening. Data presented includes all post-baseline treatment emergent Induction Period and MP toxicities, as well as LTFP toxicities for those participants who did not enter the extension period. Number of participants with post-Baseline adverse events by maximum toxicity Grade have been presented.
Time Frame: Up to an average of 59 weeks
Population: Safety Maintenance Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Any AE with maximum toxicity Grade 1 | 31 | 25 | 19
  Any AE with maximum toxicity Grade 2 | 67 | 72 | 29
  Any AE with maximum toxicity Grade 3 | 15 | 14 | 3
  Any AE with maximum toxicity Grade 4 | 2 | 2 | 1

6. Primary Outcome: Number of Participants With Maximum Post-Baseline Emergent Toxicities for Clinical Chemistry Parameters
Description: Clinical chemistry parameters aspartate amino transferase (AST), alanine amino transferase (ALT), alkaline phosphatase (ALP), carbon dioxide(CO2) content/bicarbonate (HCO3), cholesterol, creatine kinase (CK), glucose, low density lipoprotein (LDL) cholesterol, lipase, potassium, and sodium, total bilirubin (TBIL) and triglycerides were evaluated. Toxicity was graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening. Data presented includes all post-baseline treatment emergent Induction Period and MP toxicities, as well as LTFP toxicities for those participants who did not enter the extension period. Number of participants with any time post-baseline maximum emergent toxicities in any of the chemistry parameters have been presented.
Time Frame: Up to an average of 59 weeks
Population: Safety Maintenance Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Maximum toxicity Grade 1 | 94 | 94 | 44
  Maximum toxicity Grade 2 | 50 | 42 | 16
  Maximum toxicity Grade 3 | 15 | 20 | 10
  Maximum toxicity Grade 4 | 10 | 7 | 2

7. Primary Outcome: Number of Participants With Maximum Post-Baseline Emergent Toxicities for Hematology Parameters
Description: Hematology parameters hemoglobin, platelet count, total neutrophils and white blood cell count were evaluated. Toxicity was graded according to DAIDS grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening. Data presented includes all post-baseline treatment emergent Induction Period and MP toxicities, as well as LTFP toxicities for those participants who did not enter the extension period. Number of participants with any time post-baseline maximum emergent toxicities in any of the hematology parameters have been presented.
Time Frame: Up to an average of 59 weeks
Population: Safety Maintenance Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Maximum toxicity Grade 1 | 23 | 17 | 7
  Maximum toxicity Grade 2 | 2 | 4 | 2
  Maximum toxicity Grade 3 | 0 | 0 | 2
  Maximum toxicity Grade 4 | 0 | 3 | 0

8. Primary Outcome: Number of Participants With Post-Baseline Urinalysis Dipstick Results
Description: Urinalysis dipstick included urine occult blood, urine glucose, urine ketones, urine nitrite, urine protein and urine leukocyte. The dipstick test gives results in a semi-quantitative manner and results for urinalysis parameters can be read as positive, trace, 1+, 2+ and 3+ indicating proportional concentrations in the urine sample. Data presented includes all post-baseline dipstick results during Induction and Maintenance Periods, as well as LTFP for those participants who did not enter the extension period.
Time Frame: Up to an average of 59 weeks
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 20 | 20 | 10
Participants
  Urine Occult Blood, Trace, n=10,11,4: number analyzed (Participants) | 10 | 11 | 4
  Urine Occult Blood, Trace, n=10,11,4 | 5 | 6 | 1
  Urine Occult Blood, 1+, n=10,11,4: number analyzed (Participants) | 10 | 11 | 4
  Urine Occult Blood, 1+, n=10,11,4 | 3 | 3 | 2
  Urine Occult Blood, 2+, n=10,11,4: number analyzed (Participants) | 10 | 11 | 4
  Urine Occult Blood, 2+, n=10,11,4 | 0 | 0 | 0
  Urine Occult Blood, 3+, n=10,11,4: number analyzed (Participants) | 10 | 11 | 4
  Urine Occult Blood, 3+, n=10,11,4 | 2 | 2 | 1
  Urine Occult Blood, Positive, n=10,11,4: number analyzed (Participants) | 10 | 11 | 4
  Urine Occult Blood, Positive, n=10,11,4 | 0 | 0 | 0
  Urine Glucose, Trace, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Urine Glucose, Trace, n=1,1,1 | 1 | 0 | 0
  Urine Glucose, 1+, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Urine Glucose, 1+, n=1,1,1 | 0 | 0 | 1
  Urine Glucose, 2+, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Urine Glucose, 2+, n=1,1,1 | 0 | 1 | 0
  Urine Glucose, 3+, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Urine Glucose, 3+, n=1,1,1 | 0 | 0 | 0
  Urine Glucose, Positive, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Urine Glucose, Positive, n=1,1,1 | 0 | 0 | 0
  Urine Ketones, Trace, n=16,20,10: number analyzed (Participants) | 16 | 20 | 10
  Urine Ketones, Trace, n=16,20,10 | 12 | 17 | 8
  Urine Ketones, 1+, n=16,20,10: number analyzed (Participants) | 16 | 20 | 10
  Urine Ketones, 1+, n=16,20,10 | 4 | 3 | 2
  Urine Ketones, 2+, n=16,20,10: number analyzed (Participants) | 16 | 20 | 10
  Urine Ketones, 2+, n=16,20,10 | 0 | 0 | 0
  Urine Ketones, 3+, n=16,20,10: number analyzed (Participants) | 16 | 20 | 10
  Urine Ketones, 3+, n=16,20,10 | 0 | 0 | 0
  Urine Ketones, Positive, n=16,20,10: number analyzed (Participants) | 16 | 20 | 10
  Urine Ketones, Positive, n=16,20,10 | 0 | 0 | 0
  Urine Nitrite, Trace, n=1,3,1: number analyzed (Participants) | 1 | 3 | 1
  Urine Nitrite, Trace, n=1,3,1 | 0 | 0 | 0
  Urine Nitrite, 1+, n=1,3,1: number analyzed (Participants) | 1 | 3 | 1
  Urine Nitrite, 1+, n=1,3,1 | 0 | 0 | 0
  Urine Nitrite, 2+, n=1,3,1: number analyzed (Participants) | 1 | 3 | 1
  Urine Nitrite, 2+, n=1,3,1 | 0 | 0 | 0
  Urine Nitrite, 3+, n=1,3,1: number analyzed (Participants) | 1 | 3 | 1
  Urine Nitrite, 3+, n=1,3,1 | 0 | 0 | 0
  Urine Nitrite, Positive, n=1,3,1: number analyzed (Participants) | 1 | 3 | 1
  Urine Nitrite, Positive, n=1,3,1 | 1 | 3 | 1
  Urine Protein, Trace, n=17,17,7: number analyzed (Participants) | 17 | 17 | 7
  Urine Protein, Trace, n=17,17,7 | 15 | 11 | 2
  Urine Protein, 1+, n=17,17,7: number analyzed (Participants) | 17 | 17 | 7
  Urine Protein, 1+, n=17,17,7 | 2 | 4 | 5
  Urine Protein, 2+, n=17,17,7: number analyzed (Participants) | 17 | 17 | 7
  Urine Protein, 2+, n=17,17,7 | 0 | 2 | 0
  Urine Protein, 3+, n=17,17,7: number analyzed (Participants) | 17 | 17 | 7
  Urine Protein, 3+, n=17,17,7 | 0 | 0 | 0
  Urine Protein, Positive, n=17,17,7: number analyzed (Participants) | 17 | 17 | 7
  Urine Protein, Positive, n=17,17,7 | 0 | 0 | 0
  Urine Leukocyte, Trace, n=20,20,8: number analyzed (Participants) | 20 | 20 | 8
  Urine Leukocyte, Trace, n=20,20,8 | 8 | 10 | 3
  Urine Leukocyte, 1+, n=20,20,8: number analyzed (Participants) | 20 | 20 | 8
  Urine Leukocyte, 1+, n=20,20,8 | 7 | 8 | 3
  Urine Leukocyte, 2+, n=20,20,8: number analyzed (Participants) | 20 | 20 | 8
  Urine Leukocyte, 2+, n=20,20,8 | 4 | 0 | 1
  Urine Leukocyte, 3+, n=20,20,8: number analyzed (Participants) | 20 | 20 | 8
  Urine Leukocyte, 3+, n=20,20,8 | 1 | 2 | 1
  Urine Leukocyte, Positive, n=20,20,8: number analyzed (Participants) | 20 | 20 | 8
  Urine Leukocyte, Positive, n=20,20,8 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <200 c/mL and <50 c/mL, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Percentage of participants with HIV-1 RNA <200 c/mL and <50 c/mL for oral dose of CAB 30 mg plus ABC/3TC during Induction Period was obtained using FDA Snapshot algorithm. The algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as well as participants who switch their concomitant ART prior to the visit of interest, as non-responders. The Intent-to-Treat Exposed (ITT-E) Population consisted of all randomized participants who received at least one dose of investigational product.
Time Frame: Week -20, Week -16, Week -12, Week -8, Week -4, Day 1
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Percentage of participants
  HIV-1 RNA<50 c/mL, Week -20 | 0
  HIV-1 RNA<50 c/mL, Week -16 | 72
  HIV-1 RNA<50 c/mL, Week -12 | 90
  HIV-1 RNA<50 c/mL, Week -8 | 89
  HIV-1 RNA<50 c/mL, Week -4 | 92
  HIV-1 RNA<50 c/mL, Day 1 | 91
  HIV-1 RNA<200 c/mL, Week -20 | 0
  HIV-1 RNA<200 c/mL, Week -16 | 94
  HIV-1 RNA<200 c/mL, Week -12 | 97
  HIV-1 RNA<200 c/mL, Week -8 | 96
  HIV-1 RNA<200 c/mL, Week -4 | 94
  HIV-1 RNA<200 c/mL, Day 1 | 94

10. Secondary Outcome: Absolute Values of Plasma HIV-1 RNA, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Plasma samples for quantitative HIV-1 RNA were collected at indicated time points. Log10 values for HIV-1 RNA have been presented.
Time Frame: Week -20, Week -16, Week -12, Week -8, Week -4, Day 1
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Log10 copies per milliliter
  Week -20, n=309 | 4.43 (0.672)
  Week -16, n=304: number analyzed (Participants) | 304
  Week -16, n=304 | 1.71 (0.229)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | 1.62 (0.108)
  Week -8, n=299: number analyzed (Participants) | 299
  Week -8, n=299 | 1.63 (0.281)
  Week -4, n=294: number analyzed (Participants) | 294
  Week -4, n=294 | 1.61 (0.080)
  Day 1, n=291: number analyzed (Participants) | 291
  Day 1, n=291 | 1.60 (0.070)

11. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Plasma samples for quantitative HIV-1 RNA were collected at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as: HIV-1 RNA(log 10) at post-baseline visit minus HIV-1 RNA(log 10) at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
Log10 copies per milliliter
  Week -16, n=304 | -2.72 (0.572)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | -2.80 (0.640)
  Week -8, n=299: number analyzed (Participants) | 299
  Week -8, n=299 | -2.79 (0.665)
  Week -4, n=294: number analyzed (Participants) | 294
  Week -4, n=294 | -2.81 (0.647)
  Day 1, n=291: number analyzed (Participants) | 291
  Day 1, n=291 | -2.82 (0.645)

12. Secondary Outcome: Absolute Values of Cluster of Differentiation 4+ (CD4+), for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Blood samples were collected at specified time points to assess CD4+ using flow cytometry. Mean and standard deviation values for CD4+ are presented.
Time Frame: Week -20, Week -16, Week -12, Week -4, Day 1
Population: ITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Cells per cubic millimeter
  Week -20, n=309 | 498.9 (180.67)
  Week -16, n=304: number analyzed (Participants) | 304
  Week -16, n=304 | 630.5 (235.09)
  Week -12, n=300: number analyzed (Participants) | 300
  Week -12, n=300 | 664.2 (256.57)
  Week -4, n=292: number analyzed (Participants) | 292
  Week -4, n=292 | 702.3 (269.60)
  Day 1, n=291: number analyzed (Participants) | 291
  Day 1, n=291 | 690.9 (261.63)

13. Secondary Outcome: Change From Baseline in CD4+, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -4, Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
Cells per cubic millimeter
  Week -16, n=304 | 131.7 (172.69)
  Week -12, n=300: number analyzed (Participants) | 300
  Week -12, n=300 | 164.5 (174.61)
  Week -4, n=292: number analyzed (Participants) | 292
  Week -4, n=292 | 201.5 (195.53)
  Day 1, n=291: number analyzed (Participants) | 291
  Day 1, n=291 | 188.7 (186.69)

14. Secondary Outcome: Number of Participants With AEs by Their Severity Grades, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events were evaluated by the investigator and graded according to the DAIDS toxicity grading, where Grade 1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening. The higher the grade, the more severe the symptoms. Number of participants with adverse events by maximum grade have been presented.
Time Frame: Up to 20 Weeks
Population: Safety Maintenance Population. It consisted of all participants who entered the Maintenance period and received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 56
Participants
  Maximum toxicity Grade 1 | 27
  Maximum toxicity Grade 2 | 15
  Maximum toxicity Grade 3 | 2
  Maximum toxicity Grade 4 | 1

15. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Toxicities for Hematology Parameters, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Hematology parameters hemoglobin, platelet count, total neutrophils and white blood cell count were evaluated. Laboratory toxicities were graded according to DAIDS grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening. Number of participants with any time post-baseline maximum emergent toxicities in any of the hematology parameters have been presented.
Time Frame: Up to Week 20
Population: Safety Population. It consists of all enrolled subjects who received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Participants
  Maximum toxicity Grade 1 | 26
  Maximum toxicity Grade 2 | 4
  Maximum toxicity Grade 3 | 1
  Maximum toxicity Grade 4 | 3

16. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Toxicities for Clinical Chemistry Parameters, for Oral Dose of CAB 30 mg Plus ABC/3TC (Induction Period)
Description: Clinical chemistry parameters AST, ALT, ALP, CO2/HCO3, cholesterol, CK, glucose, LDL cholesterol, lipase, potassium, and sodium, total TBIL and triglycerides were evaluated. Laboratory toxicities were graded according to DAIDS grading criteria, where Grade 1-mild, Grade 2-moderate, Grade 3-severe, Grade 4-potentially life-threatening. Number of participants with any time post-baseline maximum emergent toxicities in any of the chemistry parameters have been presented.
Time Frame: Up to 20 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 309
Participants
  Maximum toxicity Grade 1 | 130
  Maximum toxicity Grade 2 | 50
  Maximum toxicity Grade 3 | 16
  Maximum toxicity Grade 4 | 5

17. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP, AST and CK (Induction Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALT, ALP, AST and CK at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 306
International Units per Liter (IU/L)
  ALT, Week -16, n=306 | 0.4 (33.1)
  ALT, Week -12, n=301: number analyzed (Participants) | 301
  ALT, Week -12, n=301 | -1.3 (14.1)
  ALT, Week -8, n=297: number analyzed (Participants) | 297
  ALT, Week -8, n=297 | -0.5 (16.6)
  ALT, Week -4, n=292: number analyzed (Participants) | 292
  ALT, Week -4, n=292 | 1.5 (50.3)
  ALT, Day 1, n=287: number analyzed (Participants) | 287
  ALT, Day 1, n=287 | -1.2 (18.0)
  ALP, Week -16, n=306 | -2.1 (12.0)
  ALP, Week -12, n=301: number analyzed (Participants) | 301
  ALP, Week -12, n=301 | -2.6 (11.0)
  ALP, Week -8, n=297: number analyzed (Participants) | 297
  ALP, Week -8, n=297 | -1.2 (13.0)
  ALP, Week -4, n=292: number analyzed (Participants) | 292
  ALP, Week -4, n=292 | 0.1 (15.4)
  ALP, Day 1, n=287: number analyzed (Participants) | 287
  ALP, Day 1, n=287 | 0.1 (14.1)
  AST, Week -16, n=306 | 0.3 (33.4)
  AST, Week -12, n=301: number analyzed (Participants) | 301
  AST, Week -12, n=301 | -2.2 (13.1)
  AST, Week -8, n=296: number analyzed (Participants) | 296
  AST, Week -8, n=296 | -1.7 (15.8)
  AST, Week -4, n=292: number analyzed (Participants) | 292
  AST, Week -4, n=292 | -0.0 (30.9)
  AST, Day 1, n=286: number analyzed (Participants) | 286
  AST, Day 1, n=286 | -1.0 (25.9)
  CK, Week -16, n=306 | 19.0 (345.6)
  CK, Week -12, n=301: number analyzed (Participants) | 301
  CK, Week -12, n=301 | 29.4 (485.4)
  CK, Week -8, n=297: number analyzed (Participants) | 297
  CK, Week -8, n=297 | 26.3 (529.6)
  CK, Week -4, n=292: number analyzed (Participants) | 292
  CK, Week -4, n=292 | 33.2 (434.2)
  CK, Day 1, n=287: number analyzed (Participants) | 287
  CK, Day 1, n=287 | 69.9 (1164.7)

18. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin (Induction Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Albumin at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per Liter (G/L)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 306
Grams per Liter (G/L)
  Week -16, n=306 | 0.2 (2.3)
  Week -12, n=301: number analyzed (Participants) | 301
  Week -12, n=301 | 0.7 (2.3)
  Week -8, n=297: number analyzed (Participants) | 297
  Week -8, n=297 | 1.4 (2.6)
  Week -4, n=292: number analyzed (Participants) | 292
  Week -4, n=292 | 1.7 (2.6)
  Day 1, n=287: number analyzed (Participants) | 287
  Day 1, n=287 | 1.9 (2.8)

19. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Total Bilirubin and Creatinine (Induction Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including total Bilirubin and Creatinine at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 306
Micromoles per Liter (umol/L)
  Total Bilirubin, Week -16, n=305: number analyzed (Participants) | 305
  Total Bilirubin, Week -16, n=305 | -0.6 (4.5)
  Total Bilirubin, Week -12, n=301: number analyzed (Participants) | 301
  Total Bilirubin, Week -12, n=301 | -0.9 (4.0)
  Total Bilirubin, Week -8, n=297: number analyzed (Participants) | 297
  Total Bilirubin, Week -8, n=297 | -1.0 (4.1)
  Total Bilirubin, Week -4, n=292: number analyzed (Participants) | 292
  Total Bilirubin, Week -4, n=292 | -0.5 (4.1)
  Total Bilirubin, Day 1, n=287: number analyzed (Participants) | 287
  Total Bilirubin, Day 1, n=287 | -0.3 (4.0)
  Creatinine, Week -16, n=306 | 2.6 (7.6)
  Creatinine, Week -12, n=301: number analyzed (Participants) | 301
  Creatinine, Week -12, n=301 | 1.5 (7.8)
  Creatinine, Week -8, n=297: number analyzed (Participants) | 297
  Creatinine, Week -8, n=297 | 1.6 (7.8)
  Creatinine, Week -4, n=292: number analyzed (Participants) | 292
  Creatinine, Week -4, n=292 | 3.5 (8.7)
  Creatinine, Day 1, n=287: number analyzed (Participants) | 287
  Creatinine, Day 1, n=287 | 4.6 (9.1)

20. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: CO2, Chloride, Cholesterol, Glucose, Potassium, Sodium, Triglyceride and Urea (Induction Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including total CO2, chloride, cholesterol, glucose, potassium, sodium, triglyceride and urea at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 306
Millimoles per Liter (mmol/L)
  CO2, Week -16, n=306 | 0.2 (2.4)
  CO2, Week -12, n=301: number analyzed (Participants) | 301
  CO2, Week -12, n=301 | 0.3 (2.3)
  CO2, Week -8, n=296: number analyzed (Participants) | 296
  CO2, Week -8, n=296 | 0.4 (2.3)
  CO2, Week -4, n=292: number analyzed (Participants) | 292
  CO2, Week -4, n=292 | 0.1 (2.3)
  CO2, Day 1, n=286: number analyzed (Participants) | 286
  CO2, Day 1, n=286 | -0.8 (2.6)
  Chloride, Week -16, n=306 | 0.2 (2.3)
  Chloride, Week -12, n=301: number analyzed (Participants) | 301
  Chloride, Week -12, n=301 | 0.5 (2.2)
  Chloride, Week -8, n=297: number analyzed (Participants) | 297
  Chloride, Week -8, n=297 | 0.6 (2.3)
  Chloride, Week -4, n=292: number analyzed (Participants) | 292
  Chloride, Week -4, n=292 | 0.2 (2.3)
  Chloride, Day 1, n=287: number analyzed (Participants) | 287
  Chloride, Day 1, n=287 | 0.2 (2.3)
  Cholesterol, Week -16, n=255: number analyzed (Participants) | 255
  Cholesterol, Week -16, n=255 | 0.21 (0.6)
  Cholesterol, Week -12, n=236: number analyzed (Participants) | 236
  Cholesterol, Week -12, n=236 | 0.19 (0.5)
  Cholesterol, Week -8, n=235: number analyzed (Participants) | 235
  Cholesterol, Week -8, n=235 | 0.27 (0.5)
  Cholesterol, Week -4, n=282: number analyzed (Participants) | 282
  Cholesterol, Week -4, n=282 | 0.34 (0.5)
  Cholesterol, Day 1, n=285: number analyzed (Participants) | 285
  Cholesterol, Day 1, n=285 | 0.34 (0.6)
  Glucose, Week -16, n=255: number analyzed (Participants) | 255
  Glucose, Week -16, n=255 | 0.07 (0.7)
  Glucose, Week -12, n=236: number analyzed (Participants) | 236
  Glucose, Week -12, n=236 | 0.16 (0.7)
  Glucose, Week -8, n=235: number analyzed (Participants) | 235
  Glucose, Week -8, n=235 | 0.08 (0.7)
  Glucose, Week -4, n=281: number analyzed (Participants) | 281
  Glucose, Week -4, n=281 | 0.06 (0.7)
  Glucose, Day 1, n=282: number analyzed (Participants) | 282
  Glucose, Day 1, n=282 | -0.01 (0.7)
  Potassium, Week -16, n=306 | -0.05 (0.2)
  Potassium, Week -12, n=301: number analyzed (Participants) | 301
  Potassium, Week -12, n=301 | -0.03 (0.3)
  Potassium, Week -8, n=296: number analyzed (Participants) | 296
  Potassium, Week -8, n=296 | 0.03 (0.3)
  Potassium, Week -4, n=292: number analyzed (Participants) | 292
  Potassium, Week -4, n=292 | 0.03 (0.3)
  Potassium, Day 1, n=286: number analyzed (Participants) | 286
  Potassium, Day 1, n=286 | 0.03 (0.3)
  Sodium, Week -16, n=306 | -0.1 (1.8)
  Sodium, Week -12, n=301: number analyzed (Participants) | 301
  Sodium, Week -12, n=301 | 0.1 (1.8)
  Sodium, Week -8, n=297: number analyzed (Participants) | 297
  Sodium, Week -8, n=297 | 0.2 (1.9)
  Sodium, Week -4, n=292: number analyzed (Participants) | 292
  Sodium, Week -4, n=292 | 0.4 (2.0)
  Sodium, Day 1, n=287: number analyzed (Participants) | 287
  Sodium, Day 1, n=287 | 0.3 (1.9)
  Triglyceride, Week -16, n=3: number analyzed (Participants) | 3
  Triglyceride, Week -16, n=3 | -0.69 (0.1)
  Triglyceride, Week -12, n=2: number analyzed (Participants) | 2
  Triglyceride, Week -12, n=2 | -0.37 (0.1)
  Triglyceride, Week -8, n=2: number analyzed (Participants) | 2
  Triglyceride, Week -8, n=2 | 0.29 (0.4)
  Triglyceride, Week -4, n=278: number analyzed (Participants) | 278
  Triglyceride, Week -4, n=278 | 0.20 (0.9)
  Triglyceride, Day 1, n=278: number analyzed (Participants) | 278
  Triglyceride, Day 1, n=278 | -0.00 (0.7)
  Urea, Week -16, n=306 | -0.06 (1.2)
  Urea, Week -12, n=301: number analyzed (Participants) | 301
  Urea, Week -12, n=301 | -0.08 (1.2)
  Urea, Week -8, n=297: number analyzed (Participants) | 297
  Urea, Week -8, n=297 | -0.09 (1.1)
  Urea, Week -4, n=292: number analyzed (Participants) | 292
  Urea, Week -4, n=292 | -0.12 (1.3)
  Urea, Day 1, n=287: number analyzed (Participants) | 287
  Urea, Day 1, n=287 | 0.00 (1.2)

21. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lipase (Induction Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameter: Lipase at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 306
Units per Liter (U/L)
  Week -16, n=306 | 3.3 (20.0)
  Week -12, n=301: number analyzed (Participants) | 301
  Week -12, n=301 | 0.8 (15.3)
  Week -8, n=297: number analyzed (Participants) | 297
  Week -8, n=297 | 2.8 (24.3)
  Week -4, n=292: number analyzed (Participants) | 292
  Week -4, n=292 | 2.1 (23.8)
  Day 1, n=288: number analyzed (Participants) | 288
  Day 1, n=288 | -1.2 (17.7)

22. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophil, Eosinophils, Lymphocytes, Total Neutrophils, Monocytes, Platelets Count and White Blood Cells (WBC) Count (Induction Period)
Description: Blood samples were collected for the analysis of hematology parameters: Basophil, Eosinophils, Lymphocytes, Total Neutrophils, Monocytes, Platelets count and WBC at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 303
Giga cells per Liter
  Basophils, Week -16, n=303 | 0.00 (0.016)
  Basophils, Week -12, n=298: number analyzed (Participants) | 298
  Basophils, Week -12, n=298 | 0.00 (0.019)
  Basophils, Week -8, n=297: number analyzed (Participants) | 297
  Basophils, Week -8, n=297 | 0.00 (0.015)
  Basophils, Week -4, n=290: number analyzed (Participants) | 290
  Basophils, Week -4, n=290 | 0.00 (0.016)
  Basophils, Day 1, n=290: number analyzed (Participants) | 290
  Basophils, Day 1, n=290 | 0.00 (0.019)
  Eosinophils, Week -16, n=303 | 0.01 (0.131)
  Eosinophils, Week -12, n=298: number analyzed (Participants) | 298
  Eosinophils, Week -12, n=298 | 0.01 (0.123)
  Eosinophils, Week -8, n=297: number analyzed (Participants) | 297
  Eosinophils, Week -8, n=297 | 0.02 (0.127)
  Eosinophils, Week -4, n=290: number analyzed (Participants) | 290
  Eosinophils, Week -4, n=290 | 0.02 (0.136)
  Eosinophils, Day 1, n=290: number analyzed (Participants) | 290
  Eosinophils, Day 1, n=290 | 0.03 (0.161)
  Lymphocytes, Week -16, n=303 | 0.24 (0.541)
  Lymphocytes, Week -12, n=298: number analyzed (Participants) | 298
  Lymphocytes, Week -12, n=298 | 0.28 (0.573)
  Lymphocytes, Week -8, n=297: number analyzed (Participants) | 297
  Lymphocytes, Week -8, n=297 | 0.30 (0.541)
  Lymphocytes, Week -4, n=290: number analyzed (Participants) | 290
  Lymphocytes, Week -4, n=290 | 0.30 (0.574)
  Lymphocytes, Day 1, n=290: number analyzed (Participants) | 290
  Lymphocytes, Day 1, n=290 | 0.14 (0.565)
  Monocytes, Week -16, n=303 | -0.00 (0.129)
  Monocytes, Week -12, n=298: number analyzed (Participants) | 298
  Monocytes, Week -12, n=298 | 0.00 (0.139)
  Monocytes, Week -8, n=297: number analyzed (Participants) | 297
  Monocytes, Week -8, n=297 | -0.00 (0.135)
  Monocytes, Week -4, n=290: number analyzed (Participants) | 290
  Monocytes, Week -4, n=290 | -0.00 (0.132)
  Monocytes, Day 1, n=290: number analyzed (Participants) | 290
  Monocytes, Day 1, n=290 | 0.00 (0.143)
  Platelet count, Week -16, n=302: number analyzed (Participants) | 302
  Platelet count, Week -16, n=302 | 14.4 (31.56)
  Platelet count, Week -12, n=300: number analyzed (Participants) | 300
  Platelet count, Week -12, n=300 | 18.2 (32.53)
  Platelet count, Week -8, n=297: number analyzed (Participants) | 297
  Platelet count, Week -8, n=297 | 21.1 (37.00)
  Platelet count, Week -4, n=290: number analyzed (Participants) | 290
  Platelet count, Week -4, n=290 | 23.0 (35.02)
  Platelet count, Day 1, n=290: number analyzed (Participants) | 290
  Platelet count, Day 1, n=290 | 22.2 (35.32)
  Total Neutrophils, Week -16, n=303 | 0.04 (1.185)
  Total Neutrophils, Week -12, n=298: number analyzed (Participants) | 298
  Total Neutrophils, Week -12, n=298 | 0.22 (1.391)
  Total Neutrophils, Week -8, n=297: number analyzed (Participants) | 297
  Total Neutrophils, Week -8, n=297 | 0.20 (1.286)
  Total Neutrophils, Week -4, n=290: number analyzed (Participants) | 290
  Total Neutrophils, Week -4, n=290 | 0.31 (1.429)
  Total Neutrophils, Day 1, n=290: number analyzed (Participants) | 290
  Total Neutrophils, Day 1, n=290 | 0.38 (1.515)
  WBC, Week -16, n=303 | 0.31 (1.318)
  WBC, Week -12, n=298: number analyzed (Participants) | 298
  WBC, Week -12, n=298 | 0.52 (1.522)
  WBC, Week -8, n=297: number analyzed (Participants) | 297
  WBC, Week -8, n=297 | 0.54 (1.460)
  WBC, Week -4, n=290: number analyzed (Participants) | 290
  WBC, Week -4, n=290 | 0.64 (1.594)
  WBC, Day 1, n=290: number analyzed (Participants) | 290
  WBC, Day 1, n=290 | 0.57 (1.713)

23. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit (Induction Period)
Description: Blood samples were collected for the analysis of hematology parameter: Hematocrit at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
Proportion of red blood cells in blood
  Week -16, n=304 | 0.00 (0.022)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | 0.00 (0.023)
  Week -8, n=298: number analyzed (Participants) | 298
  Week -8, n=298 | 0.00 (0.024)
  Week -4, n=290: number analyzed (Participants) | 290
  Week -4, n=290 | 0.00 (0.025)
  Day 1, n=290: number analyzed (Participants) | 290
  Day 1, n=290 | 0.00 (0.025)

24. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin (Induction Period)
Description: Blood samples were collected for the analysis of hematology parameter: Hemoglobin at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
Grams per Liter
  Week -16, n=304 | 0.8 (6.94)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | 2.0 (7.07)
  Week -8, n=298: number analyzed (Participants) | 298
  Week -8, n=298 | 2.5 (7.42)
  Week -4, n=290: number analyzed (Participants) | 290
  Week -4, n=290 | 3.3 (7.95)
  Day 1, n=290: number analyzed (Participants) | 290
  Day 1, n=290 | 3.1 (7.96)

25. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume (Induction Period)
Description: Blood samples were collected for the analysis of hematology parameter: Mean Corpuscle Volume at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
Femtoliters
  Week -16, n=304 | 1.0 (1.52)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | 2.1 (1.90)
  Week -8, n=298: number analyzed (Participants) | 298
  Week -8, n=298 | 3.1 (2.49)
  Week -4, n=290: number analyzed (Participants) | 290
  Week -4, n=290 | 4.0 (2.47)
  Day 1, n=290: number analyzed (Participants) | 290
  Day 1, n=290 | 4.4 (2.57)

26. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell Count (Induction Period)
Description: Blood samples were collected for the analysis of hematology parameter: Red Blood Cell count at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: Baseline (Week -20) and Week -16, Week -12, Week -8, Week -4, Day 1
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period)
Number analyzed (Participants) | 304
10^12 cells per Liter
  Week -16, n=304 | -0.05 (0.242)
  Week -12, n=302: number analyzed (Participants) | 302
  Week -12, n=302 | -0.07 (0.254)
  Week -8, n=298: number analyzed (Participants) | 298
  Week -8, n=298 | -0.10 (0.266)
  Week -4, n=290: number analyzed (Participants) | 290
  Week -4, n=290 | -0.10 (0.284)
  Day 1, n=290: number analyzed (Participants) | 290
  Day 1, n=290 | -0.14 (0.289)

27. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level <50 c/mL and <200 c/mL Over Week 96 (Maintenance Period)
Description: Percentage of participants with HIV-1 RNA <50 c/mL and <200 c/mL was obtained using FDA Snapshot algorithm. The algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as well as participants who switch their concomitant ART prior to the visit of interest, as non-responders.
Time Frame: From Day 1 up to Week 96
Population: ITT-ME Population
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Percentage of participants
  HIV-1 RNA<50 c/mL, Day 1 | 95 | 99 | 98
  HIV-1 RNA<50 c/mL, Week 4 | 97 | 98 | 93
  HIV-1 RNA<50 c/mL, Week 8 | 98 | 97 | 95
  HIV-1 RNA<50 c/mL, Week 12 | 96 | 97 | 98
  HIV-1 RNA<50 c/mL, Week 16 | 97 | 96 | 89
  HIV-1 RNA<50 c/mL, Week 20 | 97 | 97 | 91
  HIV-1 RNA<50 c/mL, Week 24 | 96 | 94 | 91
  HIV-1 RNA<50 c/mL, Week 28 | 90 | 92 | 86
  HIV-1 RNA<50 c/mL, Week 32 | 95 | 94 | 91
  HIV-1 RNA<50 c/mL, Week 36 | 95 | 90 | 88
  HIV-1 RNA<50 c/mL, Week 40 | 92 | 91 | 86
  HIV-1 RNA<50 c/mL, Week 44 | 93 | 90 | 88
  HIV-1 RNA<50 c/mL, Week 48 | 92 | 91 | 89
  HIV-1 RNA<50 c/mL, Week 56 | 94 | 90 | 84
  HIV-1 RNA<50 c/mL, Week 64 | 95 | 90 | 86
  HIV-1 RNA<50 c/mL, Week 72 | 95 | 90 | 88
  HIV-1 RNA<50 c/mL, Week 80 | 95 | 87 | 84
  HIV-1 RNA<50 c/mL, Week 88 | 95 | 86 | 84
  HIV-1 RNA<50 c/mL, Week 96 | 94 | 87 | 84
  HIV-1 RNA<200 c/mL, Day 1 | 100 | 100 | 98
  HIV-1 RNA<200 c/mL, Week 4 | 99 | 100 | 96
  HIV-1 RNA<200 c/mL, Week 8 | 99 | 99 | 95
  HIV-1 RNA<200 c/mL, Week 12 | 97 | 98 | 98
  HIV-1 RNA<200 c/mL, Week 16 | 98 | 98 | 93
  HIV-1 RNA<200 c/mL, Week 20 | 98 | 97 | 93
  HIV-1 RNA<200 c/mL, Week 24 | 97 | 96 | 93
  HIV-1 RNA<200 c/mL, Week 28 | 94 | 95 | 91
  HIV-1 RNA<200 c/mL, Week 32 | 97 | 95 | 91
  HIV-1 RNA<200 c/mL, Week 36 | 97 | 93 | 89
  HIV-1 RNA<200 c/mL, Week 40 | 97 | 92 | 86
  HIV-1 RNA<200 c/mL, Week 44 | 95 | 91 | 89
  HIV-1 RNA<200 c/mL, Week 48 | 97 | 92 | 89
  HIV-1 RNA<200 c/mL, Week 56 | 96 | 90 | 86
  HIV-1 RNA<200 c/mL, Week 64 | 96 | 90 | 88
  HIV-1 RNA<200 c/mL, Week 72 | 96 | 90 | 88
  HIV-1 RNA<200 c/mL, Week 80 | 96 | 88 | 84
  HIV-1 RNA<200 c/mL, Week 88 | 96 | 86 | 84
  HIV-1 RNA<200 c/mL, Week 96 | 96 | 87 | 84

28. Secondary Outcome: Number of Participants With Protocol Defined Virologic Failure at Week 32 and Week 48 (Maintenance Period)
Description: Virologic failure was defined as any of the following: (1) Non-response as indicated by a less than a 1.0 log10 c/mL decrease in plasma HIV-1 RNA after 4 weeks of starting the Induction Period, which is subsequently confirmed, unless the plasma HIV-1 RNA is < 400 c/mL; (2) Rebound as indicated by two consecutive plasma HIV-1 RNA levels >=200 c/mL after prior suppression to < 200 c/mL; (3) Rebound as indicated by two consecutive plasma HIV-1 RNA that are > 0.5 log10 c/mL increase in plasma HIV-1 RNA from the nadir value on study, where the lowest HIV-1 RNA value is >=200 c/mL.
Time Frame: At Week 32 and Week 48
Population: ITT-ME Population
Measure: Number; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Week 32 | 1 | 0 | 1
  Week 48 | 2 | 0 | 1

29. Secondary Outcome: Absolute Value of Plasma HIV-1 RNA at Week 32 and Week 96 (Maintenance Period)
Description: Plasma samples for quantitative HIV-1 RNA analysis were collected at indicated time points during Maintenance Period. Log10 values for HIV-1 RNA have been presented. SD=0.000 is defined as following: if participants analyzed at a specific timepoint have resulted same values, then SD is considered equal with 0.000.
Time Frame: At Week 32 and Week 96
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 108 | 50
Log10 copies per milliliter
  Week 32 | 1.60 (0.044) | 1.59 (0.025) | 1.61 (0.112)
  Week 96: number analyzed (Participants) | 110 | 100 | 47
  Week 96 | 1.60 (0.056) | 1.59 (0.000) | 1.59 (0.000)

30. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA at Week 32 and Week 96 (Maintenance Period)
Description: Plasma samples for quantitative HIV-1 RNA analysis were collected at indicated time points during Maintenance Period. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as: HIV-1 RNA(log 10) at post-baseline visit minus HIV-1 RNA(log 10) at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 108 | 50
Log10 copies per milliliter
  Week 32 | -2.78 (0.610) | -2.88 (0.709) | -2.73 (0.561)
  Week 96: number analyzed (Participants) | 110 | 100 | 47
  Week 96 | -2.77 (0.602) | -2.89 (0.713) | -2.77 (0.582)

31. Secondary Outcome: Absolute Value of CD4+ at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry.
Time Frame: At Week 32 and Week 96
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Cells per cubic millimeter
  Week 32 | 752.3 (318.02) | 761.3 (293.07) | 891.3 (273.32)
  Week 96: number analyzed (Participants) | 109 | 100 | 47
  Week 96 | 748.6 (253.41) | 750.0 (271.11) | 906.8 (288.77)

32. Secondary Outcome: Change From Baseline in CD4+ at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as post-baseline value minus Baseline value.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Cells per cubic millimeter
  Week 32 | 264.4 (247.84) | 263.7 (217.74) | 346.1 (219.59)
  Week 96: number analyzed (Participants) | 109 | 100 | 47
  Week 96 | 257.5 (192.25) | 270.6 (210.99) | 369.9 (226.60)

33. Secondary Outcome: Number of Participants With HIV-1 Disease Progression Over Week 32 and Week 96 (Maintenance Period)
Description: HIV-associated conditions were recorded during the study and was assessed according to the Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection in Adults. The clinical categories of HIV infection as per CDC system are class A=Asymptomatic HIV infection or lymphadenopathy or acute HIV infection; class B=symptomatic non-acquired immunodeficiency syndrome (AIDS) conditions and class C=AIDS indicator conditions. Number of participants experiencing disease progression is presented, where disease progression is defined as the progression from Baseline HIV disease status as follows: CDC class A at Baseline to CDC class C event; CDC Class B at Baseline to CDC Class C event; CDC Class C at Baseline to new CDC Class C event; and CDC class A, B or C at Baseline to death.
Time Frame: At Week 32 and Week 96
Population: ITT-ME Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  From CDC Stage 1 to CDC Stage 3 Event, Week 32 | 1 | 0 | 0
  From CDC Stage 2 to CDC Stage 3 Event, Week 32 | 0 | 0 | 0
  From CDC Stage 3 to New CDC Stage 3 Event, Week 32 | 0 | 0 | 0
  From CDC Stage 1, 2 or 3 to Death, Week 32 | 0 | 1 | 0
  From CDC Stage 1 to CDC Stage 3 Event, Week 96 | 4 | 0 | 0
  From CDC Stage 2 to CDC Stage 3 Event, Week 96 | 0 | 0 | 0
  From CDC Stage 3 to New CDC Stage 3 Event, Week 96 | 0 | 0 | 0
  From CDC Stage 1, 2 or 3 to Death, Week 96 | 0 | 1 | 0

34. Secondary Outcome: Number of Participants With AEs by Their Severity Grades Over Week 32 (Maintenance Period)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Adverse events were evaluated by the investigator and graded according to the DAIDS toxicity grading, where Grade 1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Number of participants with adverse events by maximum grade have been presented.
Time Frame: Up to Week 32
Population: Safety Maintenance Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Grade 1 | 35 | 29 | 23
  Grade 2 | 65 | 69 | 22
  Grade 3 | 14 | 13 | 1
  Grade 4 | 1 | 2 | 0

35. Secondary Outcome: Number of Participants With AEs by Their Severity Grades Over Week 96 (Maintenance Period)
Description: as for outcome 34
Time Frame: Up to Week 96
Population: Safety Maintenance Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 115 | 115 | 56
Participants
  Grade 1 | 23 | 21 | 24
  Grade 2 | 71 | 74 | 26
  Grade 3 | 19 | 18 | 4
  Grade 4 | 2 | 2 | 0

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP, AST and CK at Week 32 and Week 96 (Maintenance Period)
Description: as for outcome 17
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International Units per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
International Units per Liter
  ALT, Week 32 | -2.4 (13.4) | -2.7 (13.5) | -5.0 (19.5)
  ALP, Week 32 | -1.2 (14.6) | -3.8 (15.0) | -1.3 (11.6)
  AST, Week 32 | -2.8 (12.5) | -2.2 (14.5) | -8.3 (30.6)
  CK, Week 32 | 51.4 (651.0) | 93.4 (446.9) | 38.8 (394.9)
  ALT, Week 96: number analyzed (Participants) | 109 | 100 | 47
  ALT, Week 96 | 1.8 (19.19) | -2.2 (14.42) | -2.7 (22.17)
  ALP, Week 96: number analyzed (Participants) | 109 | 100 | 47
  ALP, Week 96 | -3.1 (15.59) | -3.4 (15.64) | -2.8 (12.34)
  AST, Week 96: number analyzed (Participants) | 109 | 100 | 47
  AST, Week 96 | -1.0 (15.45) | -4.0 (9.31) | -8.8 (32.57)
  CK, Week 96: number analyzed (Participants) | 109 | 100 | 47
  CK, Week 96 | 21.1 (490.00) | 13.7 (153.92) | -13.9 (227.98)

37. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including Albumin at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Grams per Liter
  Week 32 | 1.4 (3.0) | 0.9 (2.9) | 1.1 (2.8)
  Week 96: number analyzed (Participants) | 109 | 100 | 47
  Week 96 | 1.0 (2.76) | 0.9 (2.87) | 0.2 (2.61)

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Total Bilirubin and Creatinine at Week 32 and Week 96 (Maintenance Period)
Description: as for outcome 19
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Micromoles per Liter
  Total Bilirubin, Week 32 | 0.8 (4.4) | 0.4 (3.6) | -0.6 (4.4)
  Creatinine, Week 32 | 2.7 (8.5) | 3.8 (8.7) | 2.7 (6.1)
  Total Bilirubin, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Total Bilirubin, Week 96 | 0.0 (3.78) | -0.3 (4.11) | -1.1 (4.25)
  Creatinine, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Creatinine, Week 96 | 3.11 (8.515) | 4.27 (8.730) | 4.42 (6.105)

39. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Total CO2, Chloride, Cholesterol, Glucose, Potassium, Sodium, Triglyceride and Urea at Week 32 and Week 96 (Maintenance Period)
Description: as for outcome 20
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimoles per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Millimoles per Liter
  Total CO2, Week 32 | -0.8 (2.1) | -1.5 (2.4) | -1.1 (2.4)
  Chloride, Week 32 | -0.2 (2.2) | -0.3 (2.4) | 0.1 (2.1)
  Cholesterol, Week 32: number analyzed (Participants) | 109 | 106 | 50
  Cholesterol, Week 32 | 0.37 (0.6) | 0.47 (0.7) | 0.25 (0.5)
  Glucose, Week 32: number analyzed (Participants) | 109 | 106 | 50
  Glucose, Week 32 | 0.13 (1.0) | 0.03 (0.7) | -0.05 (0.6)
  Potassium, Week 32 | 0.01 (0.3) | -0.05 (0.3) | -0.04 (0.2)
  Sodium, Week 32 | 0.4 (2.0) | -0.1 (1.8) | 0.0 (1.7)
  Triglycerides, Week 32: number analyzed (Participants) | 107 | 105 | 50
  Triglycerides, Week 32 | 0.08 (0.9) | -0.00 (1.7) | 0.06 (0.7)
  Urea, Week 32 | 0.15 (1.3) | 0.23 (1.4) | -0.01 (1.4)
  Total CO2, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Total CO2, Week 96 | -0.8 (2.88) | -1.1 (2.64) | -0.1 (2.47)
  Chloride, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Chloride, Week 96 | -0.1 (2.32) | -0.4 (2.53) | 0.3 (2.12)
  Cholesterol, Week 96: number analyzed (Participants) | 105 | 96 | 46
  Cholesterol, Week 96 | 0.554 (0.6724) | 0.731 (0.7380) | 0.348 (0.6490)
  Glucose, Week 96: number analyzed (Participants) | 106 | 96 | 46
  Glucose, Week 96 | 0.12 (0.729) | 0.11 (0.667) | 0.02 (0.745)
  Potassium, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Potassium, Week 96 | 0.11 (0.378) | -0.04 (0.408) | -0.03 (0.314)
  Sodium, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Sodium, Week 96 | -0.1 (1.85) | -0.4 (2.07) | -0.4 (1.96)
  Triglycerides, Week 96: number analyzed (Participants) | 103 | 95 | 46
  Triglycerides, Week 96 | 0.084 (0.9000) | 0.080 (1.4964) | 0.197 (0.4972)
  Urea, Week 96: number analyzed (Participants) | 109 | 100 | 47
  Urea, Week 96 | 0.09 (1.393) | -0.01 (1.230) | 0.12 (1.461)

40. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lipase at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including Lipase at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Units per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 112 | 108 | 50
Units per Liter
  Week 32 | -1.2 (33.2) | -4.4 (15.4) | -3.9 (14.7)
  Week 96: number analyzed (Participants) | 109 | 101 | 47
  Week 96 | 3.5 (22.00) | -0.8 (14.73) | -2.3 (14.21)

41. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophil, Eosinophils, Lymphocytes, Total Neutrophils, Monocytes, Platelet Count and WBC Count at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of hematology parameters including Basophil, Eosinophils, Lymphocytes, Total Neutrophils, Monocytes, Platelet count and WBC count at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 110 | 107 | 48
10^9 cells per Liter
  Basophils, Week 32: number analyzed (Participants) | 110 | 106 | 48
  Basophils, Week 32 | 0.00 (0.012) | -0.00 (0.022) | 0.00 (0.010)
  Eosinophils, Week 32: number analyzed (Participants) | 110 | 106 | 48
  Eosinophils, Week 32 | 0.01 (0.146) | 0.23 (1.985) | -0.01 (0.143)
  Lymphocytes, Week 32: number analyzed (Participants) | 110 | 106 | 48
  Lymphocytes, Week 32 | 0.34 (0.661) | 0.26 (0.694) | 0.48 (0.635)
  Monocytes, Week 32: number analyzed (Participants) | 110 | 106 | 48
  Monocytes, Week 32 | -0.02 (0.152) | -0.03 (0.144) | -0.00 (0.144)
  Platelet count, Week 32 | 18.7 (38.28) | 20.6 (44.93) | 11.6 (33.33)
  Total Neutrophils, Week 32: number analyzed (Participants) | 110 | 106 | 48
  Total Neutrophils, Week 32 | 0.59 (1.505) | 0.34 (1.489) | 0.94 (1.365)
  WBC count, Week 32: number analyzed (Participants) | 110 | 106 | 48
  WBC count, Week 32 | 0.93 (1.670) | 0.81 (2.881) | 1.41 (1.529)
  Basophils, Week 96: number analyzed (Participants) | 110 | 101 | 48
  Basophils, Week 96 | 0.004 (0.0139) | 0.000 (0.0204) | 0.006 (0.0157)
  Eosinophils, Week 96: number analyzed (Participants) | 110 | 101 | 48
  Eosinophils, Week 96 | 0.015 (0.1461) | 0.021 (0.1013) | -0.013 (0.1528)
  Lymphocytes, Week 96: number analyzed (Participants) | 110 | 101 | 48
  Lymphocytes, Week 96 | 0.325 (0.6356) | 0.290 (0.6793) | 0.534 (0.5408)
  Monocytes, Week 96: number analyzed (Participants) | 110 | 101 | 48
  Monocytes, Week 96 | -0.009 (0.1685) | -0.014 (0.1781) | -0.005 (0.1443)
  Platelet count, Week 96: number analyzed (Participants) | 110 | 101 | 46
  Platelet count, Week 96 | 21.9 (40.07) | 21.1 (41.49) | 15.3 (39.28)
  Total Neutrophils, Week 96: number analyzed (Participants) | 110 | 101 | 48
  Total Neutrophils, Week 96 | 0.381 (1.3060) | 0.515 (1.6200) | 0.783 (1.0747)
  WBC count, Week 96: number analyzed (Participants) | 110 | 101 | 48
  WBC count, Week 96 | 0.72 (1.545) | 0.82 (1.786) | 1.31 (1.144)

42. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of hematology parameters including Hematocrit at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 107 | 48
Proportion of red blood cells in blood
  Week 32 | 0.01 (0.026) | 0.01 (0.027) | 0.01 (0.027)
  Week 96: number analyzed (Participants) | 110 | 101 | 48
  Week 96 | 0.0114 (0.02880) | 0.0134 (0.03125) | 0.0124 (0.02748)

43. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of hematology parameters including Hemoglobin at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 107 | 48
Grams per Liter
  Week 32 | 2.0 (8.56) | 0.8 (8.45) | 1.7 (8.38)
  Week 96: number analyzed (Participants) | 110 | 101 | 48
  Week 96 | 3.9 (8.95) | 4.3 (9.92) | 4.1 (8.11)

44. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of hematology parameters including Mean Corpuscle Volume at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 107 | 48
Femtoliters
  Week 32 | 2.5 (1.97) | 2.3 (2.54) | 7.1 (2.88)
  Week 96: number analyzed (Participants) | 110 | 101 | 48
  Week 96 | 0.1 (2.99) | 0.3 (2.54) | 5.3 (3.14)

45. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cell Count at Week 32 and Week 96 (Maintenance Period)
Description: Blood samples were collected for the analysis of hematology parameters including Red Blood Cell count at indicated time points. Baseline (Week -20) refers to the last available value up to and including the date of first induction period dosing with CAB 30 mg plus ABC/3TC. Change from Baseline was defined as value at post-baseline visit minus value at Baseline.
Time Frame: At Week 32 and Week 96 (compared with Baseline [Week -20])
Population: Safety Maintenance Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 111 | 107 | 48
10^12 cells per Liter
  Week 32 | 0.03 (0.286) | 0.02 (0.278) | -0.20 (0.296)
  Week 96: number analyzed (Participants) | 110 | 101 | 48
  Week 96 | 0.12 (0.294) | 0.14 (0.310) | -0.13 (0.293)

46. Secondary Outcome: Average Initial Concentration (C0) and Maximum Plasma Concentration (Cmax) of CAB LA (Q4W IM and Q8W IM Dosing) (Maintenance Period)
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of CAB LA. The PK Concentration Population included all participants who received CAB LA and/or RPV LA and underwent PK sampling during the study, and provided available CAB LA and/or RPV LA plasma concentration data.
Time Frame: Up to Week 32
Population: PK Concentration Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period)
Number analyzed (Participants) | 115 | 115
Micrograms per milliliter
  C0 | 1.43 (54) | 2.35 (32)
  Cmax | 3.55 (56) | 3.50 (39)

47. Secondary Outcome: Average Initial Concentration (C0) and Cmax of RPV LA (Q4W IM and Q8W IM Dosing) (Maintenance Period)
Description: Blood samples were collected at indicated time points for PK analysis of RPV LA. C0 and Cmax of RPV LA (Q4W IM and Q8W IM dosing) was evaluated.
Time Frame: Up to Week 32
Population: PK Concentration Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period)
Number analyzed (Participants) | 115 | 115
Nanograms per milliliter
  C0 | 49.3 (41) | 77.2 (35)
  Cmax | 104 (47) | 111 (40)

48. Secondary Outcome: Trough Concentration (Ctrough) of CAB LA (Q8W IM Dosing) Used for Assessment of Steady State (Maintenance Period)
Description: Blood samples were collected at indicated time points for PK analysis of CAB LA. Ctrough is the lowest concentration reached by a drug before the next dose is administered. Ctrough for CAB LA (Q8W IM dosing) which were considered for the assessment of steady state are presented.
Time Frame: Pre-dose on Weeks 16, 24 and 32
Population: PK Concentration Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period)
Number analyzed (Participants) | 87
Micrograms per milliliter
  Week 16, n=87 | 1.6902 (0.80471)
  Week 24, n=86: number analyzed (Participants) | 86
  Week 24, n=86 | 1.6051 (0.78254)
  Week 32, n=84: number analyzed (Participants) | 84
  Week 32, n=84 | 1.5330 (0.70822)

49. Secondary Outcome: Ctrough of CAB LA (Q4W IM Dosing) Used for Assessment of Steady State (Maintenance Period)
Description: Blood samples were collected at indicated time points for PK analysis of CAB LA. Ctrough is the lowest concentration reached by a drug before the next dose is administered. Ctrough for CAB LA (Q4W IM dosing) which were considered for the assessment of steady state are presented.
Time Frame: Pre-dose on Weeks 16, 20, 24, 28 and 32
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period)
Number analyzed (Participants) | 85
Micrograms per milliliter
  Week 16, n=78: number analyzed (Participants) | 78
  Week 16, n=78 | 2.2703 (0.92102)
  Week 20, n=77: number analyzed (Participants) | 77
  Week 20, n=77 | 2.3861 (0.76176)
  Week 24, n=78: number analyzed (Participants) | 78
  Week 24, n=78 | 2.6342 (1.29093)
  Week 28, n=82: number analyzed (Participants) | 82
  Week 28, n=82 | 2.4365 (0.86420)
  Week 32, n=85 | 2.4715 (0.89893)

50. Secondary Outcome: Ctrough of RPV LA (Q8W IM Dosing) Used for Assessment of Steady State (Maintenance Period)
Description: Blood samples were collected at indicated time points for PK analysis of RPV LA. Ctrough is the lowest concentration reached by a drug before the next dose is administered. Ctrough for RPV LA (Q8W IM dosing) which were considered for the assessment of steady state are presented.
Time Frame: Pre-dose on Weeks 16, 24 and 32
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period)
Number analyzed (Participants) | 87
Nanograms per milliliter
  Week 16, n=87 | 41.94 (17.575)
  Week 24, n=85: number analyzed (Participants) | 85
  Week 24, n=85 | 47.97 (22.341)
  Week 32, n=83: number analyzed (Participants) | 83
  Week 32, n=83 | 57.24 (22.926)

51. Secondary Outcome: Ctrough of RPV LA (Q4W IM Dosing) Used for Assessment of Steady State (Maintenance Period)
Description: Blood samples were collected at indicated time points for PK analysis of RPV LA. Ctrough is the lowest concentration reached by a drug before the next dose is administered. Ctrough for RPV LA (Q4W IM dosing) which were considered for the assessment of steady state are presented.
Time Frame: Pre-dose on Weeks 16, 20, 24, 28 and 32
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period)
Number analyzed (Participants) | 85
Nanograms per milliliter
  Week 16, n=78: number analyzed (Participants) | 78
  Week 16, n=78 | 66.92 (25.986)
  Week 20, n=77: number analyzed (Participants) | 77
  Week 20, n=77 | 74.55 (29.156)
  Week 24, n=78: number analyzed (Participants) | 78
  Week 24, n=78 | 76.84 (27.976)
  Week 28, n=83: number analyzed (Participants) | 83
  Week 28, n=83 | 80.84 (31.297)
  Week 32, n=85 | 90.34 (34.549)

52. Secondary Outcome: Pharmacodynamic Response (HIV-1 RNA<50 c/mL) in Relation With PK Parameter (AUC[0-tau]) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between pharmacodynamics response (HIV-1 RNA<50 c/mL) at Week 32 and plasma PK parameter: area under plasma concentration-time curve from time zero to the end of dosing interval (AUC [0-tau]) of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "HIV-1 RNA<50 c/mL" (success) and the independent variable is PK parameter (AUC [0-tau]). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter AUC (0-tau).
  Standard Error (SE)=0.000 is defined as following: if for all participants was resulted same value for the specific timepoint, then SE is equal with 0.000 .
Time Frame: Up to Week 32
Population: PK Concentration Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 86 | 84 | 0
Change in log odds
  CAB LA | 0.00 (0.001) | 0.00 (0.002) |
  RPV LA | 0.00 (0.000) | 0.00 (0.000) |

53. Secondary Outcome: Pharmacodynamic Response (HIV-1 RNA<50 c/mL) in Relation With PK Parameter (Average C0) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between pharmacodynamics response (HIV-1 RNA<50 c/mL) at Week 32 and plasma PK parameter: Average C0 of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "HIV-1 RNA<50 c/mL" (success) and the independent variable is PK parameter (Average C0). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter Average C0.
Time Frame: Up to Week 32
Population: as for outcome 48
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 101 | 108 | 50
Change in log odds
  CAB LA, n=100,108, 50: number analyzed (Participants) | 100 | 108 | 50
  CAB LA, n=100,108, 50 | 0.64 (0.837) | 2.39 (1.903) | 0.39 (0.528)
  RPV LA, n=101,104,49: number analyzed (Participants) | 101 | 104 | 49
  RPV LA, n=101,104,49 | 0.00 (0.025) | 0.01 (0.039) | -0.01 (0.020)

54. Secondary Outcome: Pharmacodynamic Response (HIV-1 RNA<50 c/mL) in Relation With PK Parameter (Cmax) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between pharmacodynamics response (HIV-1 RNA<50 c/mL) at Week 32 and plasma PK parameter: Cmax of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "HIV-1 RNA<50 c/mL" (success) and the independent variable is PK parameter (Cmax). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter Cmax.
Time Frame: Up to Week 32
Population: as for outcome 48
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 98 | 97 | 0
Change in log odds
  CAB LA, n=98, 97,0 | -0.01 (0.174) | 1.64 (1.707) |
  RPV LA, n=97,96,0: number analyzed (Participants) | 97 | 96 | 0
  RPV LA, n=97,96,0 | 0.00 (0.010) | 0.01 (0.027) |

55. Secondary Outcome: Virologic Failure (From MSDF Algorithm) in Relation With PK Parameter (AUC[0-tau]) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between virologic failure at Week 32 and plasma PK parameter: AUC (0-tau) of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "virologic failure" and the independent variable is PK parameter (AUC [0-tau]). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter AUC (0-tau).
  SE=0.000 is defined as following: if for all participants was resulted same value for the specific timepoint, then SE is equal with 0.000.
Time Frame: Up to Week 32
Population: PK Concentration Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 86 | 84 | 0
Change in log odds
  CAB LA | -0.00 (0.001) | -0.00 (0.002) |
  RPV LA | 0.00 (0.000) | -0.00 (0.000) |

56. Secondary Outcome: Virologic Failure (From MSDF Algorithm) in Relation With PK Parameter (Average C0) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between virologic failure at Week 32 and plasma PK parameter: Average C0 of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "virologic failure" and the independent variable is PK parameter (Average C0). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter Average C0.
Time Frame: Up to Week 32
Population: as for outcome 48
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 101 | 108 | 50
Change in log odds
  CAB LA, n=100,108, 50: number analyzed (Participants) | 100 | 108 | 50
  CAB LA, n=100,108, 50 | -1.01 (1.014) | -2.39 (1.903) | -0.53 (0.796)
  RPV LA, n=101,104,49: number analyzed (Participants) | 101 | 104 | 49
  RPV LA, n=101,104,49 | -0.00 (0.027) | -0.01 (0.039) | -0.01 (0.038)

57. Secondary Outcome: Virologic Failure (From MSDF Algorithm) in Relation With PK Parameter (Cmax) of CAB LA and RPV LA at Week 32 (Maintenance Period)
Description: Logistic regression was used to examine the correlation between virologic failure at Week 32 and plasma PK parameter: Cmax of CAB LA and RPV LA per arm using MSDF (Missing, Switch or Discontinuation = Failure) algorithm. Estimates were obtained from logistic statistical model where the dependent variable is "virologic failure" and the independent variable is PK parameter (Cmax). Slopes and standard error are presented. Estimated effect represents the change in log odds for a one-unit increase in the PK parameter Cmax.
Time Frame: Up to Week 32
Population: as for outcome 48
Measure: Mean (Standard Error); unit: Change in log odds
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 98 | 97 | 0
Change in log odds
  CAB LA, n=98, 97,0 | -0.45 (0.509) | -1.64 (1.707) |
  RPV LA, n=97,96,0: number analyzed (Participants) | 97 | 96 | 0
  RPV LA, n=97,96,0 | -0.00 (0.012) | -0.01 (0.027) |

58. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance
Description: Plasma samples were collected to assess treatment emergent Genotypic Resistance for participants who had confirmed virologic failure. Number of participants who had any Integrase Inhibitor (INI) mutations or major mutations of other classes (Nucleoside reverse transcriptase inhibitor [NRTI], Non-nucleoside reverse transcriptase inhibitor [NNRTI], protease inhibitor [PI])are presented.
Time Frame: Up to Week 32
Population: On-trt Genotypic Resistance Population consisted of all participants in the ITT-E Population with available On-treatment genotypic resistance data, at time of protocol defined virologic failure.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 1 | 0 | 1
Participants
  INI mutations | 0 |  | 0
  Major mutations of other classes | 0 |  | 0

59. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance
Description: Plasma samples were collected for drug resistance testing. Number of participants, with treatment emergent phenotypic resistance to INI, NNRTI, NRTI and/or PI were summarized. Overall susceptibility of the drug was categorized as sensitive, partially sensitive and resistant.
Time Frame: Up to Week 32
Population: On-trt Phenotypic Resistance Population consisted of all participants in the ITT-E Population with available On-treatment phynotypic resistance data, at time of protocol defined virologic failure.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 1 | 0 | 1
Participants
  INI, Sensitive | 1 |  | 1
  INI, Partially sensitive | 0 |  | 0
  INI, Resistant | 0 |  | 0
  NNRTI, Sensitive | 1 |  | 1
  NNRTI, Partially sensitive | 0 |  | 0
  NNRTI, Resistant | 0 |  | 0
  NRTI, Sensitive | 1 |  | 1
  NRTI, Partially sensitive | 0 |  | 0
  NRTI, Resistant | 0 |  | 0
  PI, Sensitive | 1 |  | 1
  PI, Partially sensitive | 0 |  | 0
  PI, Resistant | 0 |  | 0

60. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level <50 c/mL Over Week 32 by Subgroups (Maintenance Period)
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as well as participants who switch their concomitant ART prior to the visit of interest, as non-responders. Data is presented for following subgroups: Baseline plasma HIV-1 RNA levels, Baseline CD4+ cell count, Race and HIV Risk factor (Homosexual contact [HC] and not injectable drug user).
Time Frame: Up to Week 32
Population: ITT-ME Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 99 | 94 | 49
Percentage of participants
  Baseline HIV-1 RNA<100000 c/mL, n=99,87,49: number analyzed (Participants) | 99 | 87 | 49
  Baseline HIV-1 RNA<100000 c/mL, n=99,87,49 | 96 | 92 | 94
  Baseline HIV-1 RNA>=100000 c/mL, n=16,28,7: number analyzed (Participants) | 16 | 28 | 7
  Baseline HIV-1 RNA>=100000 c/mL, n=16,28,7 | 88 | 100 | 71
  Baseline HIV-1 RNA<1000 c/mL, n=0,3,1: number analyzed (Participants) | 0 | 3 | 1
  Baseline HIV-1 RNA<1000 c/mL, n=0,3,1 |  | 100 | 100
  Baseline HIV-1 RNA 1000 to<10000c/mL, n=26,25,13: number analyzed (Participants) | 26 | 25 | 13
  Baseline HIV-1 RNA 1000 to<10000c/mL, n=26,25,13 | 100 | 84 | 92
  Baseline HIV-1 RNA 1000 to <50000c/mL, n=50,42,25: number analyzed (Participants) | 50 | 42 | 25
  Baseline HIV-1 RNA 1000 to <50000c/mL, n=50,42,25 | 49 | 39 | 24
  Baseline HIV-1 RNA 50000 to<100000c/mL,n=23,17,10: number analyzed (Participants) | 23 | 17 | 10
  Baseline HIV-1 RNA 50000 to<100000c/mL,n=23,17,10 | 87 | 100 | 90
  Baseline HIV-1 RNA>=100000 to<200000c/mL,n=9,13,2: number analyzed (Participants) | 9 | 13 | 2
  Baseline HIV-1 RNA>=100000 to<200000c/mL,n=9,13,2 | 89 | 100 | 50
  Baseline plasma HIV-1 RNA >=200000 c/mL, n=7,15,5: number analyzed (Participants) | 7 | 15 | 5
  Baseline plasma HIV-1 RNA >=200000 c/mL, n=7,15,5 | 86 | 100 | 80
  Baseline CD4+ cell count <200 cells/mm^3, n=3,2,0: number analyzed (Participants) | 3 | 2 | 0
  Baseline CD4+ cell count <200 cells/mm^3, n=3,2,0 | 100 | 100 |
  Baseline CD4+ count 200 to<350cells/mm^3,n=30,23,8: number analyzed (Participants) | 30 | 23 | 8
  Baseline CD4+ count 200 to<350cells/mm^3,n=30,23,8 | 97 | 100 | 88
  Baseline CD4+ count >=350 cells/mm^3, n=82,90,48: number analyzed (Participants) | 82 | 90 | 48
  Baseline CD4+ count >=350 cells/mm^3, n=82,90,48 | 94 | 92 | 92
  Race-White, n=93,94,39: number analyzed (Participants) | 93 | 94 | 39
  Race-White, n=93,94,39 | 95 | 94 | 95
  Race-Non-White, n=22,21,17: number analyzed (Participants) | 22 | 21 | 17
  Race-Non-White, n=22,21,17 | 95 | 95 | 82
  HC and not injectable drug user, n=98,90,40: number analyzed (Participants) | 98 | 90 | 40
  HC and not injectable drug user, n=98,90,40 | 96 | 94 | 90
  No HC and not injectable drug user, n=17,25,16: number analyzed (Participants) | 17 | 25 | 16
  No HC and not injectable drug user, n=17,25,16 | 88 | 92 | 94

61. Secondary Outcome: Percentage of Participants With Protocol Defined Virologic Failure (PDVF) at Week 32 by Subgroups(Maintenance Period)
Description: Virologic failure was defined as any of the following: (1) Non-response as indicated by a less than a 1.0 log10 c/mL decrease in plasma HIV-1 RNA after 4 weeks of starting the Induction Period, which is subsequently confirmed, unless the plasma HIV-1 RNA is < 400 c/mL; (2) Rebound as indicated by two consecutive plasma HIV-1 RNA levels >=200 c/mL after prior suppression to <200 c/mL; (3) Rebound as indicated by two consecutive plasma HIV-1 RNA that are > 0.5 log10 c/mL increase in plasma HIV-1 RNA from the nadir value on study, where the lowest HIV-1 RNA value is >=200 c/mL. Data is presented for following subgroups: Baseline plasma HIV-1 RNA levels, Baseline CD4+ cell count, Race and HIV Risk factor (Homosexual contact [HC] and not injectable drug user).
Time Frame: Up to Week 32
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Number; unit: Percentage of participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 99 | 94 | 49
Percentage of participants
  Baseline HIV-1 RNA<100000 c/mL, n=99,87,49: number analyzed (Participants) | 99 | 87 | 49
  Baseline HIV-1 RNA<100000 c/mL, n=99,87,49 | 3 | 1 | 0
  Baseline HIV-1 RNA>=100000 c/mL, n=16,28,7: number analyzed (Participants) | 16 | 28 | 7
  Baseline HIV-1 RNA>=100000 c/mL, n=16,28,7 | 13 | 0 | 29
  Baseline HIV-1 RNA<1000 c/mL, n=0,3,1: number analyzed (Participants) | 0 | 3 | 1
  Baseline HIV-1 RNA<1000 c/mL, n=0,3,1 |  | 0 | 0
  Baseline HIV-1 RNA 1000 to<10000c/mL, n=26,25,13: number analyzed (Participants) | 26 | 25 | 13
  Baseline HIV-1 RNA 1000 to<10000c/mL, n=26,25,13 | 0 | 4 | 0
  Baseline HIV-1 RNA 1000 to <50000c/mL, n=50,42,25: number analyzed (Participants) | 50 | 42 | 25
  Baseline HIV-1 RNA 1000 to <50000c/mL, n=50,42,25 | 2 | 0 | 0
  Baseline HIV-1 RNA 50000 to<100000c/mL,n=23,17,10: number analyzed (Participants) | 23 | 17 | 10
  Baseline HIV-1 RNA 50000 to<100000c/mL,n=23,17,10 | 9 | 0 | 0
  Baseline HIV-1 RNA>=100000 to<200000c/mL,n=9,13,2: number analyzed (Participants) | 9 | 13 | 2
  Baseline HIV-1 RNA>=100000 to<200000c/mL,n=9,13,2 | 11 | 0 | 50
  Baseline plasma HIV-1 RNA >=200000 c/mL, n=7,15,5: number analyzed (Participants) | 7 | 15 | 5
  Baseline plasma HIV-1 RNA >=200000 c/mL, n=7,15,5 | 14 | 0 | 20
  Baseline CD4+ cell count <200 cells/mm^3, n=3,2,0: number analyzed (Participants) | 3 | 2 | 0
  Baseline CD4+ cell count <200 cells/mm^3, n=3,2,0 | 0 | 0 |
  Baseline CD4+ count 200 to<350cells/mm^3,n=30,23,8: number analyzed (Participants) | 30 | 23 | 8
  Baseline CD4+ count 200 to<350cells/mm^3,n=30,23,8 | 0 | 0 | 13
  Baseline CD4+ count >=350 cells/mm^3, n=82,90,48: number analyzed (Participants) | 82 | 90 | 48
  Baseline CD4+ count >=350 cells/mm^3, n=82,90,48 | 6 | 1 | 2
  Race-White, n=93,94,39: number analyzed (Participants) | 93 | 94 | 39
  Race-White, n=93,94,39 | 4 | 1 | 0
  Race-Non-White, n=22,21,17: number analyzed (Participants) | 22 | 21 | 17
  Race-Non-White, n=22,21,17 | 5 | 0 | 12
  HC and not injectable drug user, n=98,90,40: number analyzed (Participants) | 98 | 90 | 40
  HC and not injectable drug user, n=98,90,40 | 3 | 1 | 5
  No HC and not injectable drug user, n=17,25,16: number analyzed (Participants) | 17 | 25 | 16
  No HC and not injectable drug user, n=17,25,16 | 12 | 0 | 0

62. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Status Version (HIVTSQ[s]) Total Score at Week 32 and Week 96 (Maintenance Period)
Description: The HIVTSQ(s) was developed to evaluate treatments for HIV and participant satisfaction. It has total 14 items and each items are scored from 6 (very satisfied) to 0 (very dissatisfied). Items 1 to 12 are summed to produce the Total Treatment Satisfaction Score with a possible range of 0 to 72. Higher scores represent greater treatment satisfaction as compared to the past few weeks.
Time Frame: At Week 32 and Week 96
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 109 | 106 | 50
Scores on a scale
  Week 32 | 68.4 (4.48) | 66.6 (6.47) | 65.1 (5.83)
  Week 96: number analyzed (Participants) | 108 | 100 | 46
  Week 96 | 68.4 (4.34) | 67.0 (5.20) | 63.5 (9.75)

63. Secondary Outcome: HIV Treatment Satisfaction Questionnaire - Change Version (HIVTSQ[c]) Total Score at Week 32 (Maintenance Period)
Description: The HIVTSQ(c) was developed to evaluate treatments for HIV and participant satisfaction. It has total 14 items and each items are scored from +3 ('much more satisfied', 'much more convenient', 'much more flexible', etc.) to -3 ('much less satisfied', 'much less convenient', 'much less flexible', etc.). Items 1 to 12 (excluding Items 7b and 9b) are summed to produce a Total Treatment Satisfaction Score (change) with a possible range of -33 to +33. The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment.
Time Frame: Week 32
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 106 | 100 | 49
Scores on a scale | 30.9 (7.56) | 28.9 (8.53) | 20.5 (14.09)

64. Secondary Outcome: Number of Participants With HIV Medication Questionnaire (HIVMQ) Item E and F Scores at Week 32 (Maintenance Period)
Description: The HIVMQ was developed to assess participant reported medication adherence. It has 6 items (a, b, c, d, e, f). Item E (How often do you find it inconvenient or difficult to take/receive medication as recommended?) and Item F (How much pain/discomfort have experienced with this medication?). Each of these 2 items are scored from 0 (none of the time) to 6 (all of the time). The higher the score, the greater the adherence to medication. Number of participants with HIVMQ Item E and F Scores at Week 32 by their score categories (0: none of the time to 6: all of the time) are presented.
Time Frame: Week 32
Population: ITT-ME Population. Only those participants available at the specified time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 109 | 106 | 50
Participants
  Item E, score 0 | 80 | 73 | 16
  Item E, score 1 | 12 | 14 | 13
  Item E, score 2 | 3 | 2 | 2
  Item E, score 3 | 2 | 6 | 3
  Item E, score 4 | 0 | 1 | 1
  Item E, score 5 | 2 | 4 | 12
  Item E, score 6 | 10 | 6 | 3
  Item F, Score 0 | 40 | 33 | 29
  Item F, Score 1 | 35 | 43 | 12
  Item F, Score 2 | 17 | 16 | 2
  Item F, Score 3 | 6 | 5 | 2
  Item F, Score 4 | 7 | 3 | 3
  Item F, Score 5 | 4 | 4 | 0
  Item F, Score 6 | 0 | 2 | 2

65. Secondary Outcome: Number of Participants With HIV Medication Questionnaire (HIVMQ) Item E and F Scores at Week 96 (Maintenance Period)
Description: The HIVMQ was developed to assess participant reported medication adherence. It has 6 items (a, b, c, d, e, f). Item E (How often do you find it inconvenient or difficult to take/receive medication as recommended?) and Item F (How much pain/discomfort have experienced with this medication?). Each of these 2 items are scored from 0 (none of the time) to 6 (all of the time). The higher the score, the greater the adherence to medication. Number of participants with HIVMQ Item E and F Scores at Week 96 by their score categories (0: none of the time to 6: all of the time) are presented.
Time Frame: Week 96
Population: Analysis was performed on the participants that received exclusively an oral regimen during the 96-weeks period [CAB 30mg+ABC/3TC QD (Induction Period and Maintenance Period) group], as pre-specified in Protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period and Maintenance Period)
Number analyzed (Participants) | 46
Participants
  Item E, score 0 | 18
  Item E, score 1 | 10
  Item E, score 2 | 3
  Item E, score 3 | 2
  Item E, score 4 | 1
  Item E, score 5 | 9
  Item E, score 6 | 3
  Item F, Score 0 | 3
  Item F, Score 1 | 8
  Item F, Score 2 | 4
  Item F, Score 3 | 1
  Item F, Score 4 | 0
  Item F, Score 5 | 1
  Item F, Score 6 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected from start of the study treatment up to end of Extension and LTFU Periods (up to approximately 468 weeks).
Description: Safety population included all randomized participants who received at least one dose of study drug, based on the study phase they were included in.
Groups:
- CAB 30 mg+ABC/3TC QD: On Day 1 of the Maintenance period, participants who successfully completed the Induction period, were randomized to receive CAB and ABC/3TC QD for 96 weeks. Eligible participants had the option to continue study participation in Extension Period by switching to an optimized IM CAB LA+ RPV LA regimen of their choice (Q8W or Q4W).
Arm/Group | CAB 30 mg+ABC/3TC QD (Induction Period) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) | CAB 30 mg+ABC/3TC QD | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) | Long-Term Follow-Up Group
All-Cause Mortality (participants affected / at risk) | 1/309 | 0/115 | 3/115 | 0/56 | 0/34 | 0/10 | 0/43
Serious Adverse Events (participants affected / at risk) | 8/309 | 31/115 | 31/115 | 9/56 | 9/34 | 1/10 | 7/43
Other Adverse Events (participants affected / at risk) | 145/309 | 115/115 | 115/115 | 52/56 | 34/34 | 10/10 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB 30 mg+ABC/3TC QD (Induction Period) (N=309) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) (N=115) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) (N=115) | CAB 30 mg+ABC/3TC QD (N=56) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) (N=34) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) (N=10) | Long-Term Follow-Up Group (N=43)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine perforation (Injury, poisoning and procedural complications) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor neurone disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy alcoholic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Buried penis syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB 30 mg+ABC/3TC QD (Induction Period) (N=309) | CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Maintenance and Extension Period) (N=115) | CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Maintenance and Extension Period) (N=115) | CAB 30 mg+ABC/3TC QD (N=56) | Optimized CAB LA 600 mg+RPV LA 900 mg IM-Q8W (Extension Period) (N=34) | Optimized CAB LA 400 mg+RPV LA 600 mg IM-Q4W (Extension Period) (N=10) | Long-Term Follow-Up Group (N=43)
Injection site pain (General disorders) | 0 (0) | 111 (2749) | 114 (3533) | 0 (0) | 31 (486) | 8 (197) | 4 (4)
Injection site swelling (General disorders) | 0 (0) | 41 (209) | 43 (293) | 0 (0) | 6 (9) | 3 (3) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 46 (327) | 57 (675) | 0 (0) | 12 (34) | 5 (14) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 32 (156) | 33 (263) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 40 (285) | 40 (305) | 0 (0) | 4 (10) | 2 (3) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 32 (161) | 29 (218) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Fatigue (General disorders) | 19 (19) | 13 (14) | 19 (28) | 4 (5) | 3 (3) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 23 (33) | 20 (33) | 3 (3) | 3 (4) | 0 (0) | 3 (3)
Injection site bruising (General disorders) | 0 (0) | 24 (65) | 18 (93) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 8 (14) | 14 (19) | 9 (11) | 3 (4) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 20 (66) | 23 (122) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 10 (11) | 15 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 7 (20) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 6 (11) | 13 (69) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (27) | 54 (129) | 54 (146) | 22 (39) | 8 (11) | 5 (13) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 30 (55) | 28 (42) | 7 (9) | 9 (12) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 36 (61) | 28 (46) | 6 (7) | 4 (5) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 28 (43) | 23 (36) | 5 (5) | 8 (10) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 19 (25) | 17 (26) | 6 (6) | 6 (9) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 19 (25) | 21 (32) | 5 (5) | 6 (8) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 21 (26) | 32 (45) | 0 (0) | 7 (10) | 3 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 8 (14) | 11 (17) | 6 (8) | 2 (3) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 0 (0) | 15 (25) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 9 (9) | 16 (19) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 8 (14) | 11 (15) | 4 (4) | 3 (7) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 7 (28) | 17 (23) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 10 (23) | 12 (18) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 8 (12) | 11 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 15 (18) | 10 (11) | 3 (3) | 3 (3) | 1 (2) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 13 (19) | 7 (7) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 9 (11) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 6 (8) | 9 (11) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 6 (6) | 9 (10) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 7 (7) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 11 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 9 (11) | 12 (20) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 8 (18) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 11 (21) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 6 (8) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 0 (0) | 11 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 8 (10) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 0 (0) | 12 (29) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 8 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 34 (34) | 39 (55) | 35 (59) | 11 (13) | 4 (5) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 38 (38) | 9 (10) | 14 (25) | 9 (11) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 14 (18) | 14 (14) | 4 (5) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 8 (9) | 8 (13) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 | 13 (13) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 11 (13) | 11 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 7 (9) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 14 (17) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 11 (14) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 10 (10) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 8 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 13 (17) | 14 (19) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 27 (27) | 30 (51) | 30 (56) | 14 (19) | 3 (6) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 9 (13) | 11 (16) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 7 (12) | 7 (10) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 27 (39) | 30 (55) | 10 (12) | 8 (16) | 3 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (14) | 13 (18) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 27 (45) | 21 (34) | 4 (7) | 6 (9) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (14) | 14 (19) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (13) | 6 (8) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (9) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 | 19 (20) | 14 (15) | 4 (4) | 4 (5) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 22 (31) | 20 (24) | 4 (4) | 3 (3) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 15 (19) | 11 (15) | 5 (6) | 4 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (11) | 11 (13) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (11) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 19 (26) | 26 (39) | 7 (8) | 4 (4) | 2 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (17) | 13 (18) | 3 (4) | 4 (4) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (20) | 10 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 12 (15) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 7 (10) | 13 (17) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 11 (19) | 18 (22) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (11) | 9 (10) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 14 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 10 (12) | 10 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 11 (12) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 25 (29) | 28 (34) | 0 (0) | 9 (9) | 2 (2) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 9 (13) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 9 (9) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02120352/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02120352/SAP_001.pdf